CLINICAL TRIAL: NCT02942017
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study Evaluating the Efficacy, Safety, and Pharmacokinetics of SAGE-547 Injection in the Treatment of Adult Female Subjects With Severe Postpartum Depression and Adult Female Subjects With Moderate Postpartum Depression
Brief Title: A Study to Evaluate Safety and Efficacy of SAGE-547 in Participants With Moderate Postpartum Depression (547-PPD-202C)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 547-PPD-202 C
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Results first posted 2019-06-13 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2022-01

CONDITIONS: Postpartum Depression
Keywords: Moderate Postpartum Depression; SAGE-547
MeSH Terms: conditions — Depression, Postpartum | interventions — brexanolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received an infusion rate equivalent to the 90 micrograms per kilogram per hour (μg/kg/h) group.
  Interventions: Drug: Placebo
- SAGE-547 90 μg/kg/h (Experimental): Participants received a 4-hour dose titration period of 30 μg/kg/h (0 to 4 hours), then 60 μg/kg/h (4 to 24 hours), then 90 μg/kg/h (24 to 52 hours), followed by a taper to 60 μg/kg/h (52 to 56 hours), and 30 μg/kg/h (56 to 60 hours).
  Interventions: Drug: SAGE-547 90 μg/kg/h

INTERVENTIONS:
Drug: Placebo — Intravenous infusion of matching placebo for SAGE-547.
  Arms: Placebo
Drug: SAGE-547 90 μg/kg/h — Intravenous infusion of SAGE-547
  Arms: SAGE-547 90 μg/kg/h

SUMMARY:
The purpose of this study was to determine if SAGE-547 Injection infused intravenously at up to 90 μg/kg/h for 60 hours reduces depressive symptoms in participants with moderate postpartum depression (PPD) compared to placebo injection as assessed by the change from baseline in Hamilton Rating Scale for Depression (HAM-D) total score.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant either must have ceased lactating at screening; or if still lactating or actively breastfeeding at screening, agreed to temporarily cease giving breastmilk to their infant(s).
* Participant had a major depressive episode that began no earlier than the third trimester and no later than the first 4 weeks following delivery, as diagnosed by Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I).
* Participant had a HAM-D total score of ≥20 and ≤25 at screening and Day 1 (prior to dosing).
* Participant was ≤ six months postpartum.
* Participant was amenable to intravenous therapy.

Key Exclusion Criteria:

* Active psychosis.
* Attempted suicide associated with index case of postpartum depression.
* Medical history of bipolar disorder.

Note: Other protocol-defined inclusion/exclusion criteria applied.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female participants between 18 and 45 years of age with PPD, defined as those who had a major depressive episode that began no earlier than the third trimester and no later than the first four weeks following delivery, as diagnosed by Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders (DSM), 4th Edition Axis I Disorders (SCID-I), a HAM-D total score of ≥20 and ≤25 at screening and Day 1 (prior to dosing), and who were ≤6 months postpartum at screening were eligible for enrollment.
Enrollment: 108 (Actual)
Dates: Start 2016-07; Primary Completion 2017-09-17 (Actual); Study Completion 2017-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Colquhoun, MD, Study Director — Sage Therapeutics
Locations (31):
- United States (31):
  - Sage Investigational Site, Chandler, Arizona
  - Sage Investigational Site, Rogers, Arkansas
  - Sage Investigational Site, Lemon Grove, California
  - Sage Investigational Site, Orange, California
  - Sage Investigational Site, Ventura, California
  - Sage Investigational Site, Gainesville, Florida
  - Sage Investigational Site, Miami, Florida
  - Sage Investigational Site, Miramar, Florida
  - Sage Investigational Site, Orlando, Florida
  - Sage Investigational Site, Pensacola, Florida
  - Sage Investigational Site, Pinellas Park, Florida
  - Sage Investigational Site, Atlanta, Georgia
  - Sage Investigational Site, Hoffman Estates, Illinois
  - Sage Investigational Site, Wichita, Kansas
  - Sage Investigational Site, Edgewood, Kentucky
  - Sage Investigational Site, Owensboro, Kentucky
  - Sage Investigational Site, Boston, Massachusetts
  - Sage Investigational Site, Flowood, Mississippi
  - Sage Investigational Site, Marlton, New Jersey
  - Sage Investigational Site, Glen Oaks, New York
  - Sage Investigational Site, Chapel Hill, North Carolina
  - Sage Investigational Site, Charlotte, North Carolina
  - Sage Investigational Site, Raleigh, North Carolina
  - Sage Investigational Site, Columbus, Ohio
  - Sage Investigational Site, Dayton, Ohio
  - Sage Investigational Site, Philadelphia, Pennsylvania
  - Sage Investigational Site, Baytown, Texas
  - Sage Investigational Site, Houston, Texas
  - Sage Investigational Site, Richardson, Texas
  - Sage Investigational Site, San Antonio, Texas
  - Sage Investigational Site, Orem, Utah

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.

REFERENCES:
- [Derived] Gerbasi ME, Meltzer-Brody S, Acaster S, Fridman M, Bonthapally V, Hodgkins P, Kanes SJ, Eldar-Lissai A. Brexanolone in Postpartum Depression: Post Hoc Analyses to Help Inform Clinical Decision-Making. J Womens Health (Larchmt). 2021 Mar;30(3):385-392. doi: 10.1089/jwh.2020.8483. Epub 2020 Nov 12. PMID 33181049
- [Derived] Meltzer-Brody S, Colquhoun H, Riesenberg R, Epperson CN, Deligiannidis KM, Rubinow DR, Li H, Sankoh AJ, Clemson C, Schacterle A, Jonas J, Kanes S. Brexanolone injection in post-partum depression: two multicentre, double-blind, randomised, placebo-controlled, phase 3 trials. Lancet. 2018 Sep 22;392(10152):1058-1070. doi: 10.1016/S0140-6736(18)31551-4. Epub 2018 Aug 31. Erratum In: Lancet. 2018 Sep 29;392(10153):1116. doi: 10.1016/S0140-6736(18)32288-8. PMID 30177236
- See also: Related Info — http://www.sagerx.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 32 centers in United States from 25 July 2016 to 11 October 2017.
Pre-assignment Details: A total of 108 participants were randomized into the study to receive either placebo or SAGE-547, 104 of whom received the study drug.
Period: Overall Study
Arm/Group | Placebo | SAGE-547 90 μg/kg/h
Started | 54 | 54
Treated | 53 | 51
Completed | 52 | 48
Not Completed | 2 | 6
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Randomized but not dosed | 1 | 3

BASELINE CHARACTERISTICS:
Population: Participants who received the study drug.
Groups:
- Placebo: Participants received an infusion rate equivalent to the 90 μg/kg/h group.
- Total: Total of all reporting groups
Arm/Group | Placebo | SAGE-547 90 μg/kg/h | Total
Number analyzed (Participants) | 53 | 51 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (5.90) | 28.2 (6.09) | 27.8 (5.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 51 | 104
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 19 | 22 | 41
  White | 33 | 29 | 62
  Other | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latina | 14 | 10 | 24
  Not Hispanic or Latina | 39 | 41 | 80
Hamilton Rating Scale for Depression (HAMD) Total Score [Mean (Standard Deviation); unit: score on a scale] — The HAM-D Total Score comprises a sum of the 17 individual item scores. Items scored in a range of 0 to 2 include: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following items are scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The Total Score can range from 0 to 52, and higher scores indicate a greater degree of depression.
  score on a scale | 22.7 (1.59) | 22.6 (1.56) | 22.7 (1.57)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at 60 Hours in 17-Item Hamilton Rating Scale for Depression (HAM-D) Total Score
Description: The HAM-D Total Score comprises a sum of the 17 individual item scores. Items scored in a range of 0 to 2 include: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following items are scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The Total Score can range from 0 to 52, and higher scores indicate a greater degree of depression. Higher scores indicate a greater degree of depression. A negative change from baseline indicates less depression. A positive change from baseline indicates more depression.
Time Frame: Baseline, Hour 60
Population: All randomized participants who started study drug infusion, had a valid baseline HAM-D assessment and at least one post-baseline HAM-D assessment. Overall number of participants analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 52 | 49
score on a scale | -12.12 (0.773) | -14.62 (0.782)
Statistical Analysis 1: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Mixed effect model for repeated measures (MMRM) was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0160, MMRM; Least Square (LS) Mean Difference = -2.50, 95% CI 2-sided [-4.52 to -0.48], Standard Error of Mean 1.019

2. Secondary Outcome: Change From Baseline in HAM-D Total Score at Day 30
Description: as for outcome 1
Time Frame: Baseline, Day 30
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 52 | 48
score on a scale | -15.23 (0.934) | -14.69 (0.955)
Statistical Analysis 1: Comparison: Placebo vs SAGE-547 90 μg/kg/h; MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6710, MMRM; LS Mean Difference = 0.54, 95% CI 2-sided [-1.98 to 3.07], Standard Error of Mean 1.271

3. Secondary Outcome: Change From Baseline in HAM-D Total Score
Description: as for outcome 1
Time Frame: Baseline, Hours 2, 4, 8, 12, 24, 36, 48, 72, and Days 7, 14 and 21
Population: All randomized participants who started study drug infusion, had a valid baseline HAM-D assessment and at least one post-baseline HAM-D assessment. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 53 | 51
score on a scale
  Change at Hour 2 | -4.00 (0.598) | -4.60 (0.595)
  Change at Hour 4 | -6.55 (0.701) | -7.32 (0.702)
  Change at Hour 8 | -7.44 (0.738) | -8.38 (0.740)
  Change at Hour 12: number analyzed (Participants) | 52 | 50
  Change at Hour 12 | -7.96 (0.758) | -9.10 (0.762)
  Change at Hour 24: number analyzed (Participants) | 53 | 50
  Change at Hour 24 | -9.81 (0.820) | -11.42 (0.827)
  Change at Hour 36: number analyzed (Participants) | 53 | 49
  Change at Hour 36 | -10.45 (0.833) | -12.31 (0.843)
  Change at Hour 48: number analyzed (Participants) | 53 | 49
  Change at Hour 48 | -10.59 (0.860) | -13.00 (0.873)
  Change at Hour 72: number analyzed (Participants) | 53 | 49
  Change at Hour 72 | -11.83 (0.829) | -15.31 (0.841)
  Change at Day 7: number analyzed (Participants) | 53 | 50
  Change at Day 7 | -10.74 (1.042) | -13.98 (1.061)
  Change at Day 14: number analyzed (Participants) | 33 | 31
  Change at Day 14 | -11.40 (0.989) | -13.43 (1.013)
  Change at Day 21: number analyzed (Participants) | 33 | 32
  Change at Day 21 | -13.26 (1.022) | -13.59 (1.041)
Statistical Analysis 1: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Hour 2: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4216, MMRM; LS Mean Difference = -0.60, 95% CI 2-sided [-2.06 to 0.87], Standard Error of Mean 0.738
Statistical Analysis 2: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Hour 4: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3947, MMRM; LS Mean Difference = -0.77, 95% CI 2-sided [-2.57 to 1.02], Standard Error of Mean 0.905
Statistical Analysis 3: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Hour 8: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3280, MMRM; LS Mean Difference = -0.95, 95% CI 2-sided [-2.86 to 0.96], Standard Error of Mean 0.962
Statistical Analysis 4: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Hour 12: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2522, MMRM; LS Mean Difference = -1.14, 95% CI 2-sided [-3.12 to 0.83], Standard Error of Mean 0.994
Statistical Analysis 5: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Hour 24: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1431, MMRM; LS Mean Difference = -1.61, 95% CI 2-sided [-3.78 to 0.55], Standard Error of Mean 1.091
Statistical Analysis 6: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Hour 36: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0991, MMRM; LS Mean Difference = -1.85, 95% CI 2-sided [-4.06 to 0.36], Standard Error of Mean 1.113
Statistical Analysis 7: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Hour 48: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0389, MMRM; LS Mean Difference = -2.42, 95% CI 2-sided [-4.71 to -0.13], Standard Error of Mean 1.155
Statistical Analysis 8: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Hour 72: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0022, MMRM; LS Mean Difference = -3.48, 95% CI 2-sided [-5.67 to -1.28], Standard Error of Mean 1.108
Statistical Analysis 9: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Day 7: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0255, MMRM; LS Mean Difference = -3.24, 95% CI 2-sided [-6.08 to -0.40], Standard Error of Mean 1.429
Statistical Analysis 10: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Day 14: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1375, MMRM; LS Mean Difference = -2.03, 95% CI 2-sided [-4.73 to 0.66], Standard Error of Mean 1.356
Statistical Analysis 11: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Day 21: MMRM was used for analysis. The change from baseline in HAM-D total score at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.8170, MMRM; LS Mean Difference = -0.33, 95% CI 2-sided [-3.11 to 2.46], Standard Error of Mean 1.400

4. Secondary Outcome: Percentage of Participants With HAM-D Response
Description: The HAM-D response is defined as having a 50% or greater reduction from baseline in HAM-D total score. The HAM-D Total Score comprises a sum of the 17 individual item scores. Items scored in a range of 0 to 2 include: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following items are scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The Total Score can range from 0 to 52, and higher scores indicate a greater degree of depression. Higher scores indicate a greater degree of depression. A negative change from baseline indicates less depression. A positive change from baseline indicates more depression.
Time Frame: Hour 60, Days 7 and 30
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 53 | 51
percentage of participants
  Hour 60: number analyzed (Participants) | 52 | 49
  Hour 60 | 59.6 | 75.5
  Day 7: number analyzed (Participants) | 53 | 50
  Day 7 | 50.9 | 66.0
  Day 30: number analyzed (Participants) | 52 | 48
  Day 30 | 78.8 | 70.8
Statistical Analysis 1: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Hour 60: Generalized estimating equation (GEE) method was used for analysis. The HAM-D response at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model; Test type: Superiority; p = 0.0168, GEE method; Odds Ratio (OR) = 2.9, 95% CI 2-sided [1.2 to 6.7]
Statistical Analysis 2: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Day 7: GEE method was used for analysis. The HAM-D response at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model; Test type: Superiority; p = 0.0482, GEE method; Odds Ratio (OR) = 2.6, 95% CI 2-sided [1.0 to 6.6]
Statistical Analysis 3: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Day 30: GEE method was used for analysis. The HAM-D response at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. An exchangeable working correlation structure is assumed for the model parameters estimation; Test type: Superiority; p = 0.5857, GEE method; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.3 to 2.0]

5. Secondary Outcome: Percentage of Participants With HAM-D Remission
Description: HAM-D remission is defined as having a HAM-D total score of ≤7. The HAM-D Total Score comprises a sum of the 17 individual item scores. Items scored in a range of 0 to 2 include: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following items are scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. The Total Score can range from 0 to 52, and higher scores indicate a greater degree of depression. Higher scores indicate a greater degree of depression. A negative change from baseline indicates less depression. A positive change from baseline indicates more depression.
Time Frame: Hour 60, Days 7 and 30
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 53 | 51
percentage of participants
  Hour 60: number analyzed (Participants) | 52 | 49
  Hour 60 | 38.5 | 61.2
  Day 7: number analyzed (Participants) | 53 | 50
  Day 7 | 32.1 | 56.0
  Day 30: number analyzed (Participants) | 52 | 48
  Day 30 | 61.5 | 47.9
Statistical Analysis 1: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Hour 60: GEE method was used for analysis. The HAM-D remission at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model; Test type: Superiority; p = 0.0033, GEE method — Hour 60:; Odds Ratio (OR) = 3.4, 95% CI 2-sided [1.5 to 7.9]
Statistical Analysis 2: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Day 7: GEE method was used for analysis. The HAM-D remission at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model; Test type: Superiority; p = 0.0046, GEE method; Odds Ratio (OR) = 3.7, 95% CI 2-sided [1.5 to 9.3]
Statistical Analysis 3: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Day 30: GEE method was used for analysis. The HAM-D remission at each visit was the dependent variable. Treatment, baseline HAM-D total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model; Test type: Superiority; p = 0.3085, GEE method; Odds Ratio (OR) = 0.6, 95% CI 2-sided [0.3 to 1.5]

6. Secondary Outcome: Change From Baseline in HAM-D Bech 6 Subscale
Description: The HAM-D Bech 6 subscale score is calculated as the sum of the following six items: Item # 1 (depressed mood), Item # 2 (feelings of guilt), Item # 7 (work and activities), Item # 8 (retardation), Item # 10 (anxiety psychic), and Item # 13 (general somatic symptoms). Each item is scored in a range of 0 to 2 or 0 to 4, with higher scores indicating a greater degree of depression. The scores were transformed to a 100-point scale with a higher score indicating a greater degree of depression. A negative change from baseline indicates less depression. A positive change from baseline indicates more depression.
Time Frame: Baseline, Hour 60, Days 7 and 30
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 53 | 51
score on a scale
  Change at Hour 60: number analyzed (Participants) | 52 | 49
  Change at Hour 60 | -29.23 (2.248) | -37.59 (2.276)
  Change at Day 7: number analyzed (Participants) | 53 | 50
  Change at Day 7 | -25.05 (2.624) | -34.80 (2.668)
  Change at Day 30: number analyzed (Participants) | 52 | 48
  Change at Day 30 | -36.24 (2.345) | -34.86 (2.390)
Statistical Analysis 1: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Hour 60: MMRM was used for analysis. The change from baseline in HAM-D subscales at each visit was the dependent variable. Treatment, baseline HAM-D subscales, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0063, MMRM; LS mean difference = -8.35, 95% CI 2-sided [-14.29 to -2.42], Standard Error of Mean 2.989
Statistical Analysis 2: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Day 7: MMRM was used for analysis. The change from baseline in HAM-D subscales at each visit was the dependent variable. Treatment, baseline HAM-D subscales, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0074, MMRM; LS mean difference = -9.75, 95% CI 2-sided [-16.83 to -2.68], Standard Error of Mean 3.566
Statistical Analysis 3: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Day 30: MMRM was used for analysis. The change from baseline in HAM-D subscales at each visit was the dependent variable. Treatment, baseline HAM-D subscales, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6637, MMRM; LS mean difference = 1.37, 95% CI 2-sided [-4.88 to 7.63], Standard Error of Mean 3.149

7. Secondary Outcome: Change From Baseline in HAM-D Individual Item Scores
Description: The HAM-D comprises individual ratings of the following symptoms scored in a range of 0 to 2: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. The following symptoms are scored in a range of 0 to 4: agitation, depressed mood, feelings of guilt, suicide, work and activities, retardation, anxiety (psychic and somatic), and hypochondriasis. Higher scores indicate a greater degree of depression. A negative change from baseline indicates less depression. A positive change from baseline indicates more depression.
Time Frame: Baseline, Hours 2, 4, 8, 12, 24, 36, 48, 60, 72, and Days 7, 14, 21, and 30
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 53 | 51
score on a scale
  Depressed Mood, Change at Hour 2 | -0.35 (0.121) | -0.45 (0.121)
  Depressed Mood, Change at Hour 4 | -0.67 (0.137) | -0.92 (0.138)
  Depressed Mood, Change at Hour 8 | -0.90 (0.136) | -1.20 (0.136)
  Depressed Mood, Change at Hour 12: number analyzed (Participants) | 52 | 50
  Depressed Mood, Change at Hour 12 | -1.05 (0.139) | -1.18 (0.140)
  Depressed Mood, Change at Hour 24: number analyzed (Participants) | 53 | 50
  Depressed Mood, Change at Hour 24 | -1.01 (0.143) | -1.34 (0.145)
  Depressed Mood, Change at Hour 36: number analyzed (Participants) | 53 | 49
  Depressed Mood, Change at Hour 36 | -1.35 (0.145) | -1.64 (0.147)
  Depressed Mood, Change at Hour 48: number analyzed (Participants) | 53 | 49
  Depressed Mood, Change at Hour 48 | -1.33 (0.144) | -1.74 (0.146)
  Depressed Mood, Change at Hour 60: number analyzed (Participants) | 52 | 49
  Depressed Mood, Change at Hour 60 | -1.62 (0.142) | -1.91 (0.144)
  Depressed Mood, Change at Hour 72: number analyzed (Participants) | 53 | 49
  Depressed Mood, Change at Hour 72 | -1.63 (0.137) | -1.93 (0.140)
  Depressed Mood, Change at Day 7: number analyzed (Participants) | 53 | 50
  Depressed Mood, Change at Day 7 | -1.43 (0.159) | -1.82 (0.161)
  Depressed Mood, Change at Day 14: number analyzed (Participants) | 33 | 31
  Depressed Mood, Change at Day 14 | -1.42 (0.170) | -1.59 (0.174)
  Depressed Mood, Change at Day 21: number analyzed (Participants) | 33 | 32
  Depressed Mood, Change at Day 21 | -1.80 (0.168) | -1.56 (0.170)
  Depressed Mood, Change at Day 30: number analyzed (Participants) | 52 | 48
  Depressed Mood, Change at Day 30 | -2.07 (0.137) | -1.89 (0.140)
  Feelings of Guilt, Change at Hour 2 | -0.37 (0.125) | -0.59 (0.125)
  Feelings of Guilt, Change at Hour 4 | -0.56 (0.127) | -1.00 (0.127)
  Feelings of Guilt, Change at Hour 8 | -0.81 (0.124) | -1.04 (0.124)
  Feelings of Guilt, Change at Hour 12: number analyzed (Participants) | 52 | 50
  Feelings of Guilt, Change at Hour 12 | -0.69 (0.127) | -0.98 (0.128)
  Feelings of Guilt, Change at Hour 24: number analyzed (Participants) | 53 | 50
  Feelings of Guilt, Change at Hour 24 | -0.86 (0.122) | -1.16 (0.123)
  Feelings of Guilt, Change at Hour 36: number analyzed (Participants) | 53 | 49
  Feelings of Guilt, Change at Hour 36 | -0.75 (0.127) | -1.09 (0.129)
  Feelings of Guilt, Change at Hour 48: number analyzed (Participants) | 53 | 49
  Feelings of Guilt, Change at Hour 48 | -0.90 (0.129) | -1.11 (0.131)
  Feelings of Guilt, Change at Hour 60: number analyzed (Participants) | 52 | 49
  Feelings of Guilt, Change at Hour 60 | -0.99 (0.119) | -1.28 (0.120)
  Feelings of Guilt, Change at Hour 72: number analyzed (Participants) | 53 | 49
  Feelings of Guilt, Change at Hour 72 | -0.94 (0.121) | -1.34 (0.123)
  Feelings of Guilt, Change at Day 7: number analyzed (Participants) | 53 | 50
  Feelings of Guilt, Change at Day 7 | -0.82 (0.135) | -1.14 (0.137)
  Feelings of Guilt, Change at Day 14: number analyzed (Participants) | 33 | 31
  Feelings of Guilt, Change at Day 14 | -0.90 (0.133) | -1.00 (0.136)
  Feelings of Guilt, Change at Day 21: number analyzed (Participants) | 33 | 32
  Feelings of Guilt, Change at Day 21 | -1.01 (0.126) | -1.11 (0.128)
  Feelings of Guilt, Change at Day 30: number analyzed (Participants) | 52 | 48
  Feelings of Guilt, Change at Day 30 | -1.31 (0.111) | -1.20 (0.112)
  Suicide, Change at Hour 2 | -0.11 (0.062) | -0.19 (0.062)
  Suicide, Change at Hour 4 | -0.20 (0.062) | -0.28 (0.062)
  Suicide, Change at Hour 8 | -0.26 (0.062) | -0.32 (0.062)
  Suicide, Change at Hour 12: number analyzed (Participants) | 52 | 50
  Suicide, Change at Hour 12 | -0.27 (0.062) | -0.36 (0.062)
  Suicide, Change at Hour 24: number analyzed (Participants) | 53 | 50
  Suicide, Change at Hour 24 | -0.31 (0.062) | -0.38 (0.062)
  Suicide, Change at Hour 36: number analyzed (Participants) | 53 | 49
  Suicide, Change at Hour 36 | -0.29 (0.062) | -0.38 (0.063)
  Suicide, Change at Hour 48: number analyzed (Participants) | 53 | 49
  Suicide, Change at Hour 48 | -0.29 (0.062) | -0.40 (0.063)
  Suicide, Change at Hour 60: number analyzed (Participants) | 52 | 49
  Suicide, Change at Hour 60 | -0.33 (0.062) | -0.40 (0.063)
  Suicide, Change at Hour 72: number analyzed (Participants) | 53 | 49
  Suicide, Change at Hour 72 | -0.33 (0.062) | -0.40 (0.063)
  Suicide, Change at Day 7: number analyzed (Participants) | 53 | 50
  Suicide, Change at Day 7 | -0.29 (0.062) | -0.30 (0.062)
  Suicide, Change at Day 14: number analyzed (Participants) | 33 | 31
  Suicide, Change at Day 14 | -0.35 (0.068) | -0.32 (0.069)
  Suicide, Change at Day 21: number analyzed (Participants) | 33 | 32
  Suicide, Change at Day 21 | -0.36 (0.068) | -0.36 (0.068)
  Suicide, Change at Day 30: number analyzed (Participants) | 52 | 48
  Suicide, Change at Day 30 | -0.37 (0.062) | -0.38 (0.063)
  Insomnia - Early, Change at Hour 2 | -0.18 (0.077) | -0.22 (0.077)
  Insomnia - Early, Change at Hour 4 | -0.35 (0.092) | -0.26 (0.092)
  Insomnia - Early, Change at Hour 8 | -0.28 (0.085) | -0.26 (0.085)
  Insomnia - Early, Change at Hour 12: number analyzed (Participants) | 52 | 50
  Insomnia - Early, Change at Hour 12 | -0.36 (0.090) | -0.25 (0.091)
  Insomnia - Early, Change at Hour 24: number analyzed (Participants) | 53 | 50
  Insomnia - Early, Change at Hour 24 | -0.54 (0.111) | -0.81 (0.113)
  Insomnia - Early, Change at Hour 36: number analyzed (Participants) | 53 | 49
  Insomnia - Early, Change at Hour 36 | -0.62 (0.115) | -0.80 (0.117)
  Insomnia - Early, Change at Hour 48: number analyzed (Participants) | 53 | 49
  Insomnia - Early, Change at Hour 48 | -0.62 (0.122) | -0.94 (0.125)
  Insomnia - Early, Change at Hour 60: number analyzed (Participants) | 52 | 49
  Insomnia - Early, Change at Hour 60 | -0.87 (0.130) | -0.96 (0.133)
  Insomnia - Early, Change at Hour 72: number analyzed (Participants) | 53 | 49
  Insomnia - Early, Change at Hour 72 | -0.54 (0.119) | -0.93 (0.122)
  Insomnia - Early, Change at Day 7: number analyzed (Participants) | 53 | 50
  Insomnia - Early, Change at Day 7 | -0.69 (0.130) | -0.95 (0.133)
  Insomnia - Early, Change at Day 14: number analyzed (Participants) | 33 | 31
  Insomnia - Early, Change at Day 14 | -0.78 (0.142) | -0.98 (0.145)
  Insomnia - Early, Change at Day 21: number analyzed (Participants) | 33 | 32
  Insomnia - Early, Change at Day 21 | -0.98 (0.156) | -0.95 (0.157)
  Insomnia - Early, Change at Day 30: number analyzed (Participants) | 52 | 48
  Insomnia - Early, Change at Day 30 | -1.05 (0.126) | -0.96 (0.130)
  Insomnia - Middle, Change at Hour 2 | -0.18 (0.089) | -0.08 (0.089)
  Insomnia - Middle, Change at Hour 4 | -0.20 (0.092) | -0.22 (0.092)
  Insomnia - Middle, Change at Hour 8 | -0.28 (0.092) | -0.22 (0.092)
  Insomnia - Middle, Change at Hour 12: number analyzed (Participants) | 52 | 50
  Insomnia - Middle, Change at Hour 12 | -0.30 (0.094) | -0.15 (0.094)
  Insomnia - Middle, Change at Hour 24: number analyzed (Participants) | 53 | 50
  Insomnia - Middle, Change at Hour 24 | -0.52 (0.103) | -0.84 (0.105)
  Insomnia - Middle, Change at Hour 36: number analyzed (Participants) | 53 | 49
  Insomnia - Middle, Change at Hour 36 | -0.64 (0.103) | -0.91 (0.105)
  Insomnia - Middle, Change at Hour 48: number analyzed (Participants) | 53 | 49
  Insomnia - Middle, Change at Hour 48 | -0.58 (0.106) | -0.88 (0.109)
  Insomnia - Middle, Change at Hour 60: number analyzed (Participants) | 52 | 49
  Insomnia - Middle, Change at Hour 60 | -0.67 (0.099) | -0.96 (0.101)
  Insomnia - Middle, Change at Hour 72: number analyzed (Participants) | 53 | 49
  Insomnia - Middle, Change at Hour 72 | -0.77 (0.101) | -1.00 (0.103)
  Insomnia - Middle, Change at Day 7: number analyzed (Participants) | 53 | 50
  Insomnia - Middle, Change at Day 7 | -0.67 (0.112) | -0.89 (0.114)
  Insomnia - Middle, Change at Day 14: number analyzed (Participants) | 33 | 31
  Insomnia - Middle, Change at Day 14 | -0.62 (0.135) | -0.85 (0.137)
  Insomnia - Middle, Change at Day 21: number analyzed (Participants) | 33 | 32
  Insomnia - Middle, Change at Day 21 | -0.81 (0.139) | -0.79 (0.138)
  Insomnia - Middle, Change at Day 30: number analyzed (Participants) | 52 | 48
  Insomnia - Middle, Change at Day 30 | -0.84 (0.120) | -0.91 (0.123)
  Insomnia - Late, Change at Hour 2 | -0.14 (0.091) | -0.03 (0.092)
  Insomnia - Late, Change at Hour 4 | -0.20 (0.095) | -0.13 (0.096)
  Insomnia - Late, Change at Hour 8 | -0.20 (0.090) | -0.23 (0.090)
  Insomnia - Late, Change at Hour 12: number analyzed (Participants) | 52 | 50
  Insomnia - Late, Change at Hour 12 | -0.21 (0.091) | -0.23 (0.092)
  Insomnia - Late, Change at Hour 24: number analyzed (Participants) | 53 | 50
  Insomnia - Late, Change at Hour 24 | -0.54 (0.100) | -0.59 (0.101)
  Insomnia - Late, Change at Hour 36: number analyzed (Participants) | 53 | 49
  Insomnia - Late, Change at Hour 36 | -0.46 (0.102) | -0.45 (0.105)
  Insomnia - Late, Change at Hour 48: number analyzed (Participants) | 53 | 49
  Insomnia - Late, Change at Hour 48 | -0.56 (0.097) | -0.61 (0.100)
  Insomnia - Late, Change at Hour 60: number analyzed (Participants) | 52 | 49
  Insomnia - Late, Change at Hour 60 | -0.60 (0.098) | -0.63 (0.100)
  Insomnia - Late, Change at Hour 72: number analyzed (Participants) | 53 | 49
  Insomnia - Late, Change at Hour 72 | -0.50 (0.104) | -0.76 (0.107)
  Insomnia - Late, Change at Day 7: number analyzed (Participants) | 53 | 50
  Insomnia - Late, Change at Day 7 | -0.46 (0.100) | -0.64 (0.102)
  Insomnia - Late, Change at Day 14: number analyzed (Participants) | 33 | 31
  Insomnia - Late, Change at Day 14 | -0.27 (0.128) | -0.66 (0.130)
  Insomnia - Late, Change at Day 21: number analyzed (Participants) | 33 | 32
  Insomnia - Late, Change at Day 21 | -0.51 (0.125) | -0.64 (0.126)
  Insomnia - Late, Change at Day 30: number analyzed (Participants) | 52 | 48
  Insomnia - Late, Change at Day 30 | -0.67 (0.099) | -0.72 (0.101)
  Work and Activities, Change at Hour 2 | -0.26 (0.109) | -0.41 (0.109)
  Work and Activities, Change at Hour 4 | -0.73 (0.130) | -0.72 (0.131)
  Work and Activities, Change at Hour 8 | -0.77 (0.139) | -1.02 (0.141)
  Work and Activities, Change at Hour 12: number analyzed (Participants) | 52 | 50
  Work and Activities, Change at Hour 12 | -1.07 (0.151) | -1.18 (0.152)
  Work and Activities, Change at Hour 24: number analyzed (Participants) | 53 | 50
  Work and Activities, Change at Hour 24 | -1.34 (0.149) | -1.33 (0.151)
  Work and Activities, Change at Hour 36: number analyzed (Participants) | 53 | 49
  Work and Activities, Change at Hour 36 | -1.54 (0.146) | -1.65 (0.149)
  Work and Activities, Change at Hour 48: number analyzed (Participants) | 53 | 49
  Work and Activities, Change at Hour 48 | -1.45 (0.138) | -1.71 (0.141)
  Work and Activities, Change at Hour 60: number analyzed (Participants) | 52 | 49
  Work and Activities, Change at Hour 60 | -1.60 (0.134) | -2.04 (0.136)
  Work and Activities, Change at Hour 72: number analyzed (Participants) | 53 | 49
  Work and Activities, Change at Hour 72 | -1.68 (0.143) | -2.06 (0.146)
  Work and Activities, Change at Day 7: number analyzed (Participants) | 53 | 50
  Work and Activities, Change at Day 7 | -1.66 (0.157) | -1.94 (0.160)
  Work and Activities, Change at Day 14: number analyzed (Participants) | 33 | 31
  Work and Activities, Change at Day 14 | -1.40 (0.161) | -1.84 (0.165)
  Work and Activities, Change at Day 21: number analyzed (Participants) | 33 | 32
  Work and Activities, Change at Day 21 | -1.75 (0.174) | -1.70 (0.178)
  Work and Activities, Change at Day 30: number analyzed (Participants) | 52 | 48
  Work and Activities, Change at Day 30 | -2.04 (0.142) | -2.00 (0.145)
  Retardation, Change at Hour 2 | -0.03 (0.088) | 0.06 (0.089)
  Retardation, Change at Hour 4 | -0.20 (0.085) | 0.00 (0.086)
  Retardation, Change at Hour 8 | -0.25 (0.085) | -0.13 (0.086)
  Retardation, Change at Hour 12: number analyzed (Participants) | 52 | 50
  Retardation, Change at Hour 12 | -0.27 (0.082) | -0.29 (0.083)
  Retardation, Change at Hour 24: number analyzed (Participants) | 53 | 50
  Retardation, Change at Hour 24 | -0.18 (0.090) | -0.17 (0.092)
  Retardation, Change at Hour 36: number analyzed (Participants) | 53 | 49
  Retardation, Change at Hour 36 | -0.35 (0.082) | -0.38 (0.084)
  Retardation, Change at Hour 48: number analyzed (Participants) | 53 | 49
  Retardation, Change at Hour 48 | -0.35 (0.079) | -0.24 (0.081)
  Retardation, Change at Hour 60: number analyzed (Participants) | 52 | 49
  Retardation, Change at Hour 60 | -0.46 (0.066) | -0.55 (0.068)
  Retardation, Change at Hour 72: number analyzed (Participants) | 53 | 49
  Retardation, Change at Hour 72 | -0.48 (0.073) | -0.44 (0.075)
  Retardation, Change at Day 7: number analyzed (Participants) | 53 | 50
  Retardation, Change at Day 7 | -0.33 (0.073) | -0.55 (0.074)
  Retardation, Change at Day 14: number analyzed (Participants) | 33 | 31
  Retardation, Change at Day 14 | -0.47 (0.061) | -0.58 (0.060)
  Retardation, Change at Day 21: number analyzed (Participants) | 33 | 32
  Retardation, Change at Day 21 | -0.51 (0.070) | -0.57 (0.068)
  Retardation, Change at Day 30: number analyzed (Participants) | 52 | 48
  Retardation, Change at Day 30 | -0.54 (0.056) | -0.55 (0.058)
  Agitation, Change at Hour 2 | -0.27 (0.078) | -0.47 (0.078)
  Agitation, Change at Hour 4 | -0.42 (0.082) | -0.65 (0.082)
  Agitation, Change at Hour 8 | -0.40 (0.081) | -0.71 (0.081)
  Agitation, Change at Hour 12: number analyzed (Participants) | 52 | 50
  Agitation, Change at Hour 12 | -0.32 (0.093) | -0.62 (0.094)
  Agitation, Change at Hour 24: number analyzed (Participants) | 53 | 50
  Agitation, Change at Hour 24 | -0.52 (0.081) | -0.74 (0.083)
  Agitation, Change at Hour 36: number analyzed (Participants) | 53 | 49
  Agitation, Change at Hour 36 | -0.40 (0.092) | -0.66 (0.094)
  Agitation, Change at Hour 48: number analyzed (Participants) | 53 | 49
  Agitation, Change at Hour 48 | -0.44 (0.087) | -0.78 (0.089)
  Agitation, Change at Hour 60: number analyzed (Participants) | 52 | 49
  Agitation, Change at Hour 60 | -0.42 (0.097) | -0.64 (0.099)
  Agitation, Change at Hour 72: number analyzed (Participants) | 53 | 49
  Agitation, Change at Hour 72 | -0.37 (0.092) | -0.74 (0.094)
  Agitation, Change at Day 7: number analyzed (Participants) | 53 | 50
  Agitation, Change at Day 7 | -0.39 (0.096) | -0.65 (0.097)
  Agitation, Change at Day 14: number analyzed (Participants) | 33 | 31
  Agitation, Change at Day 14 | -0.58 (0.107) | -0.67 (0.108)
  Agitation, Change at Day 21: number analyzed (Participants) | 33 | 32
  Agitation, Change at Day 21 | -0.56 (0.112) | -0.65 (0.114)
  Agitation, Change at Day 30: number analyzed (Participants) | 52 | 48
  Agitation, Change at Day 30 | -0.60 (0.075) | -0.73 (0.077)
  Anxiety Psychic, Change at Hour 2 | -0.45 (0.126) | -0.67 (0.126)
  Anxiety Psychic, Change at Hour 4 | -0.81 (0.138) | -0.93 (0.138)
  Anxiety Psychic, Change at Hour 8 | -0.89 (0.141) | -1.05 (0.142)
  Anxiety Psychic, Change at Hour 12: number analyzed (Participants) | 52 | 50
  Anxiety Psychic, Change at Hour 12 | -0.89 (0.143) | -1.01 (0.144)
  Anxiety Psychic, Change at Hour 24: number analyzed (Participants) | 53 | 50
  Anxiety Psychic, Change at Hour 24 | -1.00 (0.140) | -1.13 (0.141)
  Anxiety Psychic, Change at Hour 36: number analyzed (Participants) | 53 | 49
  Anxiety Psychic, Change at Hour 36 | -1.06 (0.141) | -1.20 (0.143)
  Anxiety Psychic, Change at Hour 48: number analyzed (Participants) | 53 | 49
  Anxiety Psychic, Change at Hour 48 | -0.92 (0.142) | -1.24 (0.144)
  Anxiety Psychic, Change at Hour 60: number analyzed (Participants) | 52 | 49
  Anxiety Psychic, Change at Hour 60 | -0.98 (0.131) | -1.51 (0.133)
  Anxiety Psychic, Change at Hour 72: number analyzed (Participants) | 53 | 49
  Anxiety Psychic, Change at Hour 72 | -1.08 (0.135) | -1.36 (0.137)
  Anxiety Psychic, Change at Day 7: number analyzed (Participants) | 53 | 50
  Anxiety Psychic, Change at Day 7 | -0.70 (0.133) | -1.21 (0.134)
  Anxiety Psychic, Change at Day 14: number analyzed (Participants) | 33 | 31
  Anxiety Psychic, Change at Day 14 | -0.76 (0.178) | -0.82 (0.184)
  Anxiety Psychic, Change at Day 21: number analyzed (Participants) | 33 | 32
  Anxiety Psychic, Change at Day 21 | -0.94 (0.156) | -0.83 (0.158)
  Anxiety Psychic, Change at Day 30: number analyzed (Participants) | 52 | 48
  Anxiety Psychic, Change at Day 30 | -1.25 (0.138) | -1.10 (0.141)
  Anxiety Somatic, Change at Hour 2 | -0.54 (0.100) | -0.61 (0.101)
  Anxiety Somatic, Change at Hour 4 | -0.71 (0.098) | -0.81 (0.099)
  Anxiety Somatic, Change at Hour 8 | -0.62 (0.102) | -0.69 (0.103)
  Anxiety Somatic, Change at Hour 12: number analyzed (Participants) | 52 | 50
  Anxiety Somatic, Change at Hour 12 | -0.60 (0.099) | -0.87 (0.100)
  Anxiety Somatic, Change at Hour 24: number analyzed (Participants) | 53 | 50
  Anxiety Somatic, Change at Hour 24 | -0.73 (0.103) | -0.77 (0.105)
  Anxiety Somatic, Change at Hour 36: number analyzed (Participants) | 53 | 49
  Anxiety Somatic, Change at Hour 36 | -0.75 (0.098) | -0.89 (0.100)
  Anxiety Somatic, Change at Hour 48: number analyzed (Participants) | 53 | 49
  Anxiety Somatic, Change at Hour 48 | -0.79 (0.100) | -0.96 (0.103)
  Anxiety Somatic, Change at Hour 60: number analyzed (Participants) | 52 | 49
  Anxiety Somatic, Change at Hour 60 | -0.88 (0.101) | -0.95 (0.104)
  Anxiety Somatic, Change at Hour 72: number analyzed (Participants) | 53 | 49
  Anxiety Somatic, Change at Hour 72 | -0.84 (0.088) | -1.08 (0.090)
  Anxiety Somatic, Change at Day 7: number analyzed (Participants) | 53 | 50
  Anxiety Somatic, Change at Day 7 | -0.66 (0.112) | -0.92 (0.114)
  Anxiety Somatic, Change at Day 14: number analyzed (Participants) | 33 | 31
  Anxiety Somatic, Change at Day 14 | -0.85 (0.139) | -0.63 (0.139)
  Anxiety Somatic, Change at Day 21: number analyzed (Participants) | 33 | 32
  Anxiety Somatic, Change at Day 21 | -0.90 (0.119) | -1.01 (0.118)
  Anxiety Somatic, Change at Day 30: number analyzed (Participants) | 52 | 48
  Anxiety Somatic, Change at Day 30 | -0.88 (0.110) | -0.97 (0.113)
  Somatic Symptoms GI, Change at Hour 2 | -0.22 (0.091) | -0.15 (0.092)
  Somatic Symptoms GI, Change at Hour 4 | -0.33 (0.096) | -0.39 (0.096)
  Somatic Symptoms GI, Change at Hour 8 | -0.56 (0.087) | -0.37 (0.087)
  Somatic Symptoms GI, Change at Hour 12: number analyzed (Participants) | 52 | 50
  Somatic Symptoms GI, Change at Hour 12 | -0.56 (0.090) | -0.45 (0.091)
  Somatic Symptoms GI, Change at Hour 24: number analyzed (Participants) | 53 | 50
  Somatic Symptoms GI, Change at Hour 24 | -0.48 (0.083) | -0.54 (0.084)
  Somatic Symptoms GI, Change at Hour 36: number analyzed (Participants) | 53 | 49
  Somatic Symptoms GI, Change at Hour 36 | -0.60 (0.084) | -0.51 (0.086)
  Somatic Symptoms GI, Change at Hour 48: number analyzed (Participants) | 53 | 49
  Somatic Symptoms GI, Change at Hour 48 | -0.56 (0.086) | -0.59 (0.088)
  Somatic Symptoms GI, Change at Hour 60: number analyzed (Participants) | 52 | 49
  Somatic Symptoms GI, Change at Hour 60 | -0.73 (0.091) | -0.71 (0.093)
  Somatic Symptoms GI, Change at Hour 72: number analyzed (Participants) | 53 | 49
  Somatic Symptoms GI, Change at Hour 72 | -0.77 (0.081) | -0.75 (0.082)
  Somatic Symptoms GI, Change at Day 7: number analyzed (Participants) | 53 | 50
  Somatic Symptoms GI, Change at Day 7 | -0.47 (0.093) | -0.67 (0.095)
  Somatic Symptoms GI, Change at Day 14: number analyzed (Participants) | 33 | 31
  Somatic Symptoms GI, Change at Day 14 | -0.64 (0.093) | -0.79 (0.094)
  Somatic Symptoms GI, Change at Day 21: number analyzed (Participants) | 33 | 32
  Somatic Symptoms GI, Change at Day 21 | -0.61 (0.107) | -0.83 (0.108)
  Somatic Symptoms GI, Change at Day 30: number analyzed (Participants) | 52 | 48
  Somatic Symptoms GI, Change at Day 30 | -0.77 (0.085) | -0.73 (0.087)
  Somatic Symptoms General, Change at Hour 2 | -0.18 (0.081) | -0.15 (0.079)
  Somatic Symptoms General, Change at Hour 4 | -0.29 (0.095) | -0.35 (0.094)
  Somatic Symptoms General, Change at Hour 8 | -0.38 (0.094) | -0.45 (0.093)
  Somatic Symptoms General, Change at Hour 12: number analyzed (Participants) | 52 | 50
  Somatic Symptoms General, Change at Hour 12 | -0.50 (0.094) | -0.75 (0.093)
  Somatic Symptoms General, Change at Hour 24: number analyzed (Participants) | 53 | 50
  Somatic Symptoms General, Change at Hour 24 | -0.65 (0.104) | -0.73 (0.104)
  Somatic Symptoms General, Change at Hour 36: number analyzed (Participants) | 53 | 49
  Somatic Symptoms General, Change at Hour 36 | -0.55 (0.097) | -0.69 (0.098)
  Somatic Symptoms General, Change at Hour 48: number analyzed (Participants) | 53 | 49
  Somatic Symptoms General, Change at Hour 48 | -0.61 (0.101) | -0.69 (0.102)
  Somatic Symptoms General, Change at Hour 60: number analyzed (Participants) | 52 | 49
  Somatic Symptoms General, Change at Hour 60 | -0.79 (0.105) | -0.91 (0.105)
  Somatic Symptoms General, Change at Hour 72: number analyzed (Participants) | 53 | 49
  Somatic Symptoms General, Change at Hour 72 | -0.80 (0.112) | -1.05 (0.113)
  Somatic Symptoms General, Change at Day 7: number analyzed (Participants) | 53 | 50
  Somatic Symptoms General, Change at Day 7 | -0.57 (0.102) | -0.93 (0.103)
  Somatic Symptoms General, Change at Day 14: number analyzed (Participants) | 33 | 31
  Somatic Symptoms General, Change at Day 14 | -0.66 (0.118) | -0.94 (0.118)
  Somatic Symptoms General, Change at Day 21: number analyzed (Participants) | 33 | 32
  Somatic Symptoms General, Change at Day 21 | -0.82 (0.124) | -0.67 (0.123)
  Somatic Symptoms General, Change at Day 30: number analyzed (Participants) | 52 | 48
  Somatic Symptoms General, Change at Day 30 | -0.77 (0.104) | -0.86 (0.106)
  Genital Symptoms, Change at Hour 2 | -0.05 (0.052) | 0.07 (0.053)
  Genital Symptoms, Change at Hour 4 | -0.09 (0.065) | -0.01 (0.066)
  Genital Symptoms, Change at Hour 8 | -0.07 (0.070) | -0.03 (0.070)
  Genital Symptoms, Change at Hour 12: number analyzed (Participants) | 52 | 50
  Genital Symptoms, Change at Hour 12 | -0.05 (0.083) | -0.09 (0.085)
  Genital Symptoms, Change at Hour 24: number analyzed (Participants) | 53 | 50
  Genital Symptoms, Change at Hour 24 | -0.11 (0.089) | -0.13 (0.091)
  Genital Symptoms, Change at Hour 36: number analyzed (Participants) | 53 | 49
  Genital Symptoms, Change at Hour 36 | -0.18 (0.091) | -0.31 (0.094)
  Genital Symptoms, Change at Hour 48: number analyzed (Participants) | 53 | 49
  Genital Symptoms, Change at Hour 48 | -0.18 (0.092) | -0.39 (0.095)
  Genital Symptoms, Change at Hour 60: number analyzed (Participants) | 52 | 49
  Genital Symptoms, Change at Hour 60 | -0.23 (0.084) | -0.37 (0.086)
  Genital Symptoms, Change at Hour 72: number analyzed (Participants) | 53 | 49
  Genital Symptoms, Change at Hour 72 | -0.22 (0.102) | -0.59 (0.105)
  Genital Symptoms, Change at Day 7: number analyzed (Participants) | 53 | 50
  Genital Symptoms, Change at Day 7 | -0.52 (0.112) | -0.57 (0.115)
  Genital Symptoms, Change at Day 14: number analyzed (Participants) | 33 | 31
  Genital Symptoms, Change at Day 14 | -0.56 (0.149) | -0.66 (0.152)
  Genital Symptoms, Change at Day 21: number analyzed (Participants) | 33 | 32
  Genital Symptoms, Change at Day 21 | -0.67 (0.147) | -0.76 (0.149)
  Genital Symptoms, Change at Day 30: number analyzed (Participants) | 52 | 48
  Genital Symptoms, Change at Day 30 | -0.84 (0.131) | -0.62 (0.135)
  Hypochondriasis, Change at Hour 2 | -0.14 (0.077) | -0.30 (0.077)
  Hypochondriasis, Change at Hour 4 | -0.20 (0.071) | -0.28 (0.071)
  Hypochondriasis, Change at Hour 8 | -0.22 (0.073) | -0.26 (0.073)
  Hypochondriasis, Change at Hour 12: number analyzed (Participants) | 52 | 50
  Hypochondriasis, Change at Hour 12 | -0.18 (0.076) | -0.34 (0.076)
  Hypochondriasis, Change at Hour 24: number analyzed (Participants) | 53 | 50
  Hypochondriasis, Change at Hour 24 | -0.37 (0.069) | -0.32 (0.069)
  Hypochondriasis, Change at Hour 36: number analyzed (Participants) | 53 | 49
  Hypochondriasis, Change at Hour 36 | -0.25 (0.079) | -0.30 (0.080)
  Hypochondriasis, Change at Hour 48: number analyzed (Participants) | 53 | 49
  Hypochondriasis, Change at Hour 48 | -0.35 (0.075) | -0.30 (0.076)
  Hypochondriasis, Change at Hour 60: number analyzed (Participants) | 52 | 49
  Hypochondriasis, Change at Hour 60 | -0.29 (0.075) | -0.34 (0.075)
  Hypochondriasis, Change at Hour 72: number analyzed (Participants) | 53 | 49
  Hypochondriasis, Change at Hour 72 | -0.31 (0.077) | -0.36 (0.078)
  Hypochondriasis, Change at Day 7: number analyzed (Participants) | 53 | 50
  Hypochondriasis, Change at Day 7 | -0.25 (0.088) | -0.27 (0.089)
  Hypochondriasis, Change at Day 14: number analyzed (Participants) | 33 | 31
  Hypochondriasis, Change at Day 14 | -0.14 (0.102) | -0.33 (0.104)
  Hypochondriasis, Change at Day 21: number analyzed (Participants) | 33 | 32
  Hypochondriasis, Change at Day 21 | -0.30 (0.093) | -0.35 (0.094)
  Hypochondriasis, Change at Day 30: number analyzed (Participants) | 52 | 48
  Hypochondriasis, Change at Day 30 | -0.31 (0.069) | -0.40 (0.070)
  Loss of Weight, Change at Hour 2 | -0.11 (0.055) | -0.06 (0.055)
  Loss of Weight, Change at Hour 4 | -0.17 (0.063) | -0.02 (0.063)
  Loss of Weight, Change at Hour 8 | -0.19 (0.053) | -0.08 (0.053)
  Loss of Weight, Change at Hour 12: number analyzed (Participants) | 52 | 50
  Loss of Weight, Change at Hour 12 | -0.21 (0.067) | -0.02 (0.067)
  Loss of Weight, Change at Hour 24: number analyzed (Participants) | 53 | 50
  Loss of Weight, Change at Hour 24 | -0.25 (0.067) | -0.04 (0.067)
  Loss of Weight, Change at Hour 36: number analyzed (Participants) | 53 | 49
  Loss of Weight, Change at Hour 36 | -0.23 (0.066) | -0.15 (0.067)
  Loss of Weight, Change at Hour 48: number analyzed (Participants) | 53 | 49
  Loss of Weight, Change at Hour 48 | -0.23 (0.074) | -0.11 (0.076)
  Loss of Weight, Change at Hour 60: number analyzed (Participants) | 51 | 49
  Loss of Weight, Change at Hour 60 | -0.19 (0.065) | -0.19 (0.065)
  Loss of Weight, Change at Hour 72: number analyzed (Participants) | 53 | 49
  Loss of Weight, Change at Hour 72 | -0.15 (0.076) | -0.23 (0.078)
  Loss of Weight, Change at Day 7: number analyzed (Participants) | 53 | 50
  Loss of Weight, Change at Day 7 | -0.38 (0.091) | -0.18 (0.093)
  Loss of Weight, Change at Day 14: number analyzed (Participants) | 33 | 31
  Loss of Weight, Change at Day 14 | -0.44 (0.125) | -0.39 (0.127)
  Loss of Weight, Change at Day 21: number analyzed (Participants) | 33 | 32
  Loss of Weight, Change at Day 21 | -0.38 (0.130) | -0.50 (0.132)
  Loss of Weight, Change at Day 30: number analyzed (Participants) | 52 | 48
  Loss of Weight, Change at Day 30 | -0.46 (0.111) | -0.42 (0.115)
  Insight, Change at Hour 2 | 0.01 (0.034) | -0.03 (0.034)
  Insight, Change at Hour 4 | 0.01 (0.034) | -0.05 (0.034)
  Insight, Change at Hour 8 | 0.05 (0.034) | -0.03 (0.034)
  Insight, Change at Hour 12: number analyzed (Participants) | 52 | 50
  Insight, Change at Hour 12 | -0.01 (0.034) | -0.03 (0.034)
  Insight, Change at Hour 24: number analyzed (Participants) | 53 | 50
  Insight, Change at Hour 24 | 0.01 (0.034) | -0.05 (0.034)
  Insight, Change at Hour 36: number analyzed (Participants) | 53 | 49
  Insight, Change at Hour 36 | -0.01 (0.034) | -0.01 (0.034)
  Insight, Change at Hour 48: number analyzed (Participants) | 53 | 49
  Insight, Change at Hour 48 | -0.01 (0.034) | 0.01 (0.034)
  Insight, Change at Hour 60: number analyzed (Participants) | 52 | 49
  Insight, Change at Hour 60 | -0.04 (0.034) | 0.01 (0.034)
  Insight, Change at Hour 72: number analyzed (Participants) | 53 | 49
  Insight, Change at Hour 72 | -0.01 (0.034) | 0.01 (0.034)
  Insight, Change at Day 7: number analyzed (Participants) | 53 | 50
  Insight, Change at Day 7 | -0.02 (0.034) | -0.07 (0.034)
  Insight, Change at Day 14: number analyzed (Participants) | 33 | 31
  Insight, Change at Day 14 | -0.02 (0.038) | -0.02 (0.038)
  Insight, Change at Day 21: number analyzed (Participants) | 33 | 32
  Insight, Change at Day 21 | -0.02 (0.038) | -0.02 (0.038)
  Insight, Change at Day 30: number analyzed (Participants) | 52 | 48
  Insight, Change at Day 30 | -0.02 (0.034) | -0.01 (0.034)
Statistical Analysis 1: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Depressed Mood, Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5132, MMRM; LS Mean Difference = -0.10, 95% CI 2-sided [-0.41 to 0.21], Standard Error of Mean 0.154
Statistical Analysis 2: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Depressed Mood, Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1672, MMRM; LS Mean Difference = -0.25, 95% CI 2-sided [-0.61 to 0.11], Standard Error of Mean 0.181
Statistical Analysis 3: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Depressed Mood, Hour 8:MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0963, MMRM; LS Mean Difference = -0.30, 95% CI 2-sided [-0.65 to 0.05], Standard Error of Mean 0.178
Statistical Analysis 4: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Depressed Mood, Hour 12:MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4803, MMRM; LS Mean Difference = -0.13, 95% CI 2-sided [-0.49 to 0.23], Standard Error of Mean 0.183
Statistical Analysis 5: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Depressed Mood, Hour 24:MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0844, MMRM; LS Mean Difference = -0.33, 95% CI 2-sided [-0.71 to 0.05], Standard Error of Mean 0.191
Statistical Analysis 6: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Depressed Mood, Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1325, MMRM; LS Mean Difference = -0.29, 95% CI 2-sided [-0.68 to 0.09], Standard Error of Mean 0.193
Statistical Analysis 7: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Depressed Mood, Hour 48:MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0332, MMRM; LS Mean Difference = -0.41, 95% CI 2-sided [-0.79 to -0.03], Standard Error of Mean 0.192
Statistical Analysis 8: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Depressed Mood, Hour 60:MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1273, MMRM; LS Mean Difference = -0.29, 95% CI 2-sided [-0.67 to 0.08], Standard Error of Mean 0.189
Statistical Analysis 9: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Depressed Mood, Hour 72:MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1059, MMRM; LS Mean Difference = -0.30, 95% CI 2-sided [-0.66 to 0.06], Standard Error of Mean 0.182
Statistical Analysis 10: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Depressed Mood, Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0683, MMRM; LS Mean Difference = -0.40, 95% CI 2-sided [-0.82 to 0.03], Standard Error of Mean 0.215
Statistical Analysis 11: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Depressed Mood, Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4458, MMRM; LS Mean Difference = -0.18, 95% CI 2-sided [-0.64 to 0.28], Standard Error of Mean 0.232
Statistical Analysis 12: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Depressed Mood, Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2905, MMRM; LS Mean Difference = 0.24, 95% CI 2-sided [-0.21 to 0.70], Standard Error of Mean 0.228
Statistical Analysis 13: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Depressed Mood, Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3096, MMRM; LS Mean Difference = 0.19, 95% CI 2-sided [-0.18 to 0.55], Standard Error of Mean 0.182
Statistical Analysis 14: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Feeling of Guilt, Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1925, MMRM; LS Mean Difference = -0.22, 95% CI 2-sided [-0.55 to 0.11], Standard Error of Mean 0.165
Statistical Analysis 15: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Feeling of Guilt, Hour 4:MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0101, MMRM; LS Mean Difference = -0.44, 95% CI 2-sided [-0.77 to -0.11], Standard Error of Mean 0.168
Statistical Analysis 16: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Feeling of Guilt, Hour 8:MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1546, MMRM; LS Mean Difference = -0.23, 95% CI 2-sided [-0.56 to 0.09], Standard Error of Mean 0.163
Statistical Analysis 17: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Feeling of Guilt, Hour 12:MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0901, MMRM; LS Mean Difference = -0.29, 95% CI 2-sided [-0.62 to 0.05], Standard Error of Mean 0.168
Statistical Analysis 18: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Feeling of Guilt, Hour 24:MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0717, MMRM; LS Mean Difference = -0.29, 95% CI 2-sided [-0.62 to 0.03], Standard Error of Mean 0.162
Statistical Analysis 19: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Feeling of Guilt, Hour 36:MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0468, MMRM; LS Mean Difference = -0.34, 95% CI 2-sided [-0.68 to 0.00], Standard Error of Mean 0.169
Statistical Analysis 20: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Feeling of Guilt, Hour 48:MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2222, MMRM; LS Mean Difference = -0.21, 95% CI 2-sided [-0.56 to 0.13], Standard Error of Mean 0.173
Statistical Analysis 21: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Feeling of Guilt, Hour 60:MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0682, MMRM; LS Mean Difference = -0.29, 95% CI 2-sided [-0.60 to 0.02], Standard Error of Mean 0.156
Statistical Analysis 22: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Feeling of Guilt, Hour 72:MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0147, MMRM; LS Mean Difference = -0.40, 95% CI 2-sided [-0.72 to -0.08], Standard Error of Mean 0.160
Statistical Analysis 23: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Feeling of Guilt, Day 7:MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0837, MMRM; LS Mean Difference = -0.32, 95% CI 2-sided [-0.68 to 0.04], Standard Error of Mean 0.182
Statistical Analysis 24: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Feeling of Guilt, Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5828, MMRM; LS Mean Difference = -0.10, 95% CI 2-sided [-0.46 to 0.26], Standard Error of Mean 0.179
Statistical Analysis 25: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Feeling of Guilt, Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5674, MMRM; LS Mean Difference = -0.10, 95% CI 2-sided [-0.43 to 0.24], Standard Error of Mean 0.168
Statistical Analysis 26: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Feeling of Guilt, Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4613, MMRM; LS Mean Difference = 0.11, 95% CI 2-sided [-0.18 to 0.40], Standard Error of Mean 0.145
Statistical Analysis 27: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Suicide, Hour 2:MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3240, MMRM; LS Mean Difference = -0.08, 95% CI 2-sided [-0.24 to 0.08], Standard Error of Mean 0.082
Statistical Analysis 28: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Suicide, Hour 4:MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3023, MMRM; LS Mean Difference = -0.08, 95% CI 2-sided [-0.24 to 0.08], Standard Error of Mean 0.082
Statistical Analysis 29: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Suicide, Hour 8:MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4127, MMRM; LS Mean Difference = -0.07, 95% CI 2-sided [-0.23 to 0.09], Standard Error of Mean 0.082
Statistical Analysis 30: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Suicide, Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2819, MMRM; LS Mean Difference = -0.09, 95% CI 2-sided [-0.25 to 0.07], Standard Error of Mean 0.082
Statistical Analysis 31: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Suicide, Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3884, MMRM; LS Mean Difference = -0.07, 95% CI 2-sided [-0.23 to 0.09], Standard Error of Mean 0.082
Statistical Analysis 32: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Suicide, Hour 36:MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2750, MMRM; LS Mean Difference = -0.09, 95% CI 2-sided [-0.25 to 0.07], Standard Error of Mean 0.082
Statistical Analysis 33: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Suicide, Hour 48:MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1811, MMRM; LS Mean Difference = -0.11, 95% CI 2-sided [-0.27 to 0.05], Standard Error of Mean 0.082
Statistical Analysis 34: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Suicide, Hour 60:MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3854, MMRM; LS Mean Difference = -0.07, 95% CI 2-sided [-0.23 to 0.09], Standard Error of Mean 0.082
Statistical Analysis 35: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Suicide, Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3822, MMRM; LS Mean Difference = -0.07, 95% CI 2-sided [-0.23 to 0.09], Standard Error of Mean 0.082
Statistical Analysis 36: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Suicide, Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9255, MMRM; LS Mean Difference = -0.01, 95% CI 2-sided [-0.17 to 0.15], Standard Error of Mean 0.082
Statistical Analysis 37: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Suicide, Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6714, MMRM; LS Mean Difference = 0.04, 95% CI 2-sided [-0.14 to 0.22], Standard Error of Mean 0.091
Statistical Analysis 38: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Suicide, Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9838, MMRM; LS Mean Difference = 0.00, 95% CI 2-sided [-0.18 to 0.18], Standard Error of Mean 0.091
Statistical Analysis 39: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Suicide, Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.8884, MMRM; LS Mean Difference = -0.01, 95% CI 2-sided [-0.17 to 0.15], Standard Error of Mean 0.083
Statistical Analysis 40: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Early, Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6996, MMRM; LS Mean Difference = -0.04, 95% CI 2-sided [-0.23 to 0.16], Standard Error of Mean 0.097
Statistical Analysis 41: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Early, Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4426, MMRM; LS Mean Difference = 0.09, 95% CI 2-sided [-0.15 to 0.33], Standard Error of Mean 0.121
Statistical Analysis 42: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Early, Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.8743, MMRM; LS Mean Difference = 0.02, 95% CI 2-sided [-0.20 to 0.24], Standard Error of Mean 0.110
Statistical Analysis 43: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Early, Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3498, MMRM; LS Mean Difference = 0.11, 95% CI 2-sided [-0.12 to 0.35], Standard Error of Mean 0.118
Statistical Analysis 44: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Early, Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0839, MMRM; LS Mean Difference = -0.26, 95% CI 2-sided [-0.56 to 0.04], Standard Error of Mean 0.151
Statistical Analysis 45: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Early, Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2595, MMRM; LS Mean Difference = -0.18, 95% CI 2-sided [-0.49 to 0.13], Standard Error of Mean 0.157
Statistical Analysis 46: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Early, Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0560, MMRM; LS Mean Difference = -0.32, 95% CI 2-sided [-0.66 to 0.01], Standard Error of Mean 0.168
Statistical Analysis 47: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Early, Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6187, MMRM; LS Mean Difference = -0.09, 95% CI 2-sided [-0.45 to 0.27], Standard Error of Mean 0.180
Statistical Analysis 48: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Early, Hour 72 MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0187, MMRM; LS Mean Difference = -0.39, 95% CI 2-sided [-0.72 to -0.07], Standard Error of Mean 0.163
Statistical Analysis 49: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Early, Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1531, MMRM; LS Mean Difference = -0.26, 95% CI 2-sided [-0.62 to 0.10], Standard Error of Mean 0.180
Statistical Analysis 50: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Early, Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3341, MMRM; LS Mean Difference = -0.19, 95% CI 2-sided [-0.58 to 0.20], Standard Error of Mean 0.197
Statistical Analysis 51: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Early, Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.8969, MMRM; LS Mean Difference = 0.03, 95% CI 2-sided [-0.40 to 0.46], Standard Error of Mean 0.216
Statistical Analysis 52: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Early, Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5862, MMRM; LS Mean Difference = 0.10, 95% CI 2-sided [-0.25 to 0.44], Standard Error of Mean 0.174
Statistical Analysis 53: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Middle, Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3776, MMRM; LS Mean Difference = 0.10, 95% CI 2-sided [-0.13 to 0.34], Standard Error of Mean 0.117
Statistical Analysis 54: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Middle, Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9029, MMRM; LS Mean Difference = -0.01, 95% CI 2-sided [-0.26 to 0.23], Standard Error of Mean 0.121
Statistical Analysis 55: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Middle, Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6173, MMRM; LS Mean Difference = 0.06, 95% CI 2-sided [-0.18 to 0.30], Standard Error of Mean 0.121
Statistical Analysis 56: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Middle, Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2433, MMRM; LS Mean Difference = 0.15, 95% CI 2-sided [-0.10 to 0.39], Standard Error of Mean 0.124
Statistical Analysis 57: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Middle, Hour 24 MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0234, MMRM; LS Mean Difference = -0.32, 95% CI 2-sided [-0.59 to -0.04], Standard Error of Mean 0.139
Statistical Analysis 58: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Middle, Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0540, MMRM; LS Mean Difference = -0.27, 95% CI 2-sided [-0.55 to 0.00], Standard Error of Mean 0.139
Statistical Analysis 59: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Middle, Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0406, MMRM; LS Mean Difference = -0.30, 95% CI 2-sided [-0.58 to -0.01], Standard Error of Mean 0.144
Statistical Analysis 60: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Middle, Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0295, MMRM; LS Mean Difference = -0.29, 95% CI 2-sided [-0.56 to -0.03], Standard Error of Mean 0.132
Statistical Analysis 61: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Middle, Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0925, MMRM; LS Mean Difference = -0.23, 95% CI 2-sided [-0.50 to 0.04], Standard Error of Mean 0.135
Statistical Analysis 62: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Middle, Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1631, MMRM; LS Mean Difference = -0.21, 95% CI 2-sided [-0.52 to 0.09], Standard Error of Mean 0.152
Statistical Analysis 63: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Middle, Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2213, MMRM; LS Mean Difference = -0.23, 95% CI 2-sided [-0.60 to 0.14], Standard Error of Mean 0.185
Statistical Analysis 64: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Middle, Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9175, MMRM; LS Mean Difference = 0.02, 95% CI 2-sided [-0.36 to 0.39], Standard Error of Mean 0.189
Statistical Analysis 65: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Middle, Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6763, MMRM; LS Mean Difference = -0.07, 95% CI 2-sided [-0.40 to 0.26], Standard Error of Mean 0.165
Statistical Analysis 66: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Late, Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3805, MMRM; LS Mean Difference = 0.11, 95% CI 2-sided [-0.13 to 0.35], Standard Error of Mean 0.121
Statistical Analysis 67: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Late, Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6073, MMRM; LS Mean Difference = 0.07, 95% CI 2-sided [-0.19 to 0.32], Standard Error of Mean 0.127
Statistical Analysis 68: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Late, Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7848, MMRM; LS Mean Difference = -0.03, 95% CI 2-sided [-0.27 to 0.20], Standard Error of Mean 0.119
Statistical Analysis 69: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Late, Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9038, MMRM; LS Mean Difference = -0.01, 95% CI 2-sided [-0.25 to 0.23], Standard Error of Mean 0.121
Statistical Analysis 70: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Late, Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6869, MMRM; LS Mean Difference = 0.134, 95% CI 2-sided [-0.32 to 0.21], Standard Error of Mean 0.134
Statistical Analysis 71: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Late, Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9272, MMRM; LS Mean Difference = 0.01, 95% CI 2-sided [-0.26 to 0.29], Standard Error of Mean 0.139
Statistical Analysis 72: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Late, Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6931, MMRM; LS Mean Difference = -0.05, 95% CI 2-sided [-0.31 to 0.21], Standard Error of Mean 0.131
Statistical Analysis 73: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Late, Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.8262, MMRM; LS Mean Difference = -0.03, 95% CI 2-sided [-0.29 to 0.23], Standard Error of Mean 0.132
Statistical Analysis 74: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Late, Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0749, MMRM; LS Mean Difference = -0.25, 95% CI 2-sided [-0.54 to 0.03], Standard Error of Mean 0.141
Statistical Analysis 75: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Late, Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1923, MMRM; LS Mean Difference = -0.18, 95% CI 2-sided [-0.45 to 0.09], Standard Error of Mean 0.135
Statistical Analysis 76: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Late, Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0326, MMRM; LS Mean Difference = -0.38, 95% CI 2-sided [-0.73 to -0.03], Standard Error of Mean 0.176
Statistical Analysis 77: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Late, Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4440, MMRM; LS Mean Difference = -0.13, 95% CI 2-sided [-0.47 to 0.21], Standard Error of Mean 0.171
Statistical Analysis 78: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insomnia-Late, Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7057, MMRM; LS Mean Difference = -0.05, 95% CI 2-sided [-0.32 to 0.22], Standard Error of Mean 0.134
Statistical Analysis 79: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Work and Activities, Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2865, MMRM; LS Mean Difference = -0.15, 95% CI 2-sided [-0.42 to 0.13], Standard Error of Mean 0.137
Statistical Analysis 80: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Work and Activities, Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9475, MMRM; LS Mean Difference = 0.01, 95% CI 2-sided [-0.33 to 0.35], Standard Error of Mean 0.170
Statistical Analysis 81: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Work and Activities, Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1880, MMRM; LS Mean Difference = -0.25, 95% CI 2-sided [-0.61 to 0.12], Standard Error of Mean 0.185
Statistical Analysis 82: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Work and Activities, Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5950, MMRM; LS Mean Difference = -0.11, 95% CI 2-sided [-0.51 to 0.29], Standard Error of Mean 0.203
Statistical Analysis 83: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Work and Activities, Hour 24 : MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9636, MMRM; LS Mean Difference = 0.01, 95% CI 2-sided [-0.39 to 0.41], Standard Error of Mean 0.200
Statistical Analysis 84: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Work and Activities, Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5836, MMRM; LS Mean Difference = -0.11, 95% CI 2-sided [-0.50 to 0.28], Standard Error of Mean 0.196
Statistical Analysis 85: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Work and Activities, Hour 48 : MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1568, MMRM; LS Mean Difference = -0.26, 95% CI 2-sided [-0.63 to 0.10], Standard Error of Mean 0.184
Statistical Analysis 86: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Work and Activities, Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0155, Wilcoxon (Mann-Whitney); LS Mean Difference = -0.44, 5% CI 2-sided [-0.79 to -0.09], Standard Error of Mean 0.177
Statistical Analysis 87: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Work and Activities, Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0504, MMRM; LS Mean Difference = -0.38, 95% CI 2-sided [-0.76 to 0.00], Standard Error of Mean 0.192
Statistical Analysis 88: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Work and Activities, Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1865, MMRM; LS Mean Difference = -0.28, 95% CI 2-sided [-0.70 to 0.14], Standard Error of Mean 0.212
Statistical Analysis 89: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Work and Activities, Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0518, MMRM; LS Mean Difference = -0.43, 95% CI 2-sided [-0.87 to 0.00], Standard Error of Mean 0.220
Statistical Analysis 90: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Work and Activities, Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.8330, MMRM; LS Mean Difference = 0.05, 95% CI 2-sided [-0.42 to 0.53], Standard Error of Mean 0.239
Statistical Analysis 91: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Work and Activities, Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.8440, MMRM; LS Mean Difference = 0.04, 95% CI 2-sided [-0.34 to 0.42], Standard Error of Mean 0.191
Statistical Analysis 92: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Retardation, Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4602, MMRM; LS Mean Difference = 0.09, 95% CI 2-sided [-0.15 to 0.33], Standard Error of Mean 0.121
Statistical Analysis 93: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Retardation, Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0891, MMRM; LS Mean Difference = 0.20, 95% CI 2-sided [-0.03 to 0.43], Standard Error of Mean 0.117
Statistical Analysis 94: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Retardation, Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3088, MMRM; LS Mean Difference = 0.12, 95% CI 2-sided [-0.11 to 0.35], Standard Error of Mean 0.117
Statistical Analysis 95: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Retardation, Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.8560, MMRM; LS Mean Difference = -0.02, 95% CI 2-sided [-0.24 to 0.20], Standard Error of Mean 0.112
Statistical Analysis 96: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Retardation, Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9702, MMRM; LS Mean Difference = 0.00, 95% CI 2-sided [-0.24 to 0.25], Standard Error of Mean 0.125
Statistical Analysis 97: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Retardation, Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.8001, MMRM; LS Mean Difference = -0.03, 95% CI 2-sided [-0.25 to 0.20], Standard Error of Mean 0.114
Statistical Analysis 98: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Retardation, Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3223, MMRM; LS Mean Difference = 0.11, 95% CI 2-sided [-0.11 to 0.32], Standard Error of Mean 0.109
Statistical Analysis 99: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Retardation, Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3385, MMRM; LS Mean Difference = -0.09, 95% CI 2-sided [-0.26 to 0.09], Standard Error of Mean 0.089
Statistical Analysis 100: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Retardation, Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7003, MMRM; LS Mean Difference = 0.04, 95% CI 2-sided [-0.16 to 0.24], Standard Error of Mean 0.100
Statistical Analysis 101: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Retardation, Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0311, MMRM; LS Mean Difference = -0.22, 95% CI 2-sided [-0.41 to -0.02], Standard Error of Mean 0.099
Statistical Analysis 102: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Retardation, Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1976, MMRM; LS Mean Difference = -0.10, 95% CI 2-sided [-0.26 to 0.06], Standard Error of Mean 0.079
Statistical Analysis 103: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Retardation, Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5489, MMRM; LS Mean Difference = -0.06, 95% CI 2-sided [-0.24 to 0.13], Standard Error of Mean 0.092
Statistical Analysis 104: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Retardation, Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7992, MMRM; LS Mean Difference = -0.02, 95% CI 2-sided [-0.17 to 0.13], Standard Error of Mean 0.075
Statistical Analysis 105: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Agitation, Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0573, MMRM; LS Mean Difference = -0.20, 95% CI 2-sided [-0.40 to 0.01], Standard Error of Mean 0.103
Statistical Analysis 106: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Agitation, Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0431, MMRM; LS Mean Difference = -0.22, 95% CI 2-sided [-0.44 to -0.01], Standard Error of Mean 0.110
Statistical Analysis 107: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Agitation, Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0060, MMRM; LS Mean Difference = -0.30, 95% CI 2-sided [-0.52 to -0.09], Standard Error of Mean 0.108
Statistical Analysis 108: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Agitation, Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0215, MMRM; LS Mean Difference = -0.30, 95% CI 2-sided [-0.55 to -0.04], Standard Error of Mean 0.127
Statistical Analysis 109: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Agitation, Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0422, MMRM; LS Mean Difference = -0.22, 95% CI 2-sided [-0.44 to -0.01], Standard Error of Mean 0.109
Statistical Analysis 110: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Agitation, Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0433, MMRM; LS Mean Difference = -0.26, 95% CI 2-sided [-0.51 to -0.01], Standard Error of Mean 0.126
Statistical Analysis 111: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Agitation, Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0051, MMRM; LS Mean Difference = -0.34, 95% CI 2-sided [-0.57 to -0.10], Standard Error of Mean 0.118
Statistical Analysis 112: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Agitation, Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0973, MMRM; LS Mean Difference = -0.22, 95% CI 2-sided [-0.48 to 0.04], Standard Error of Mean 0.133
Statistical Analysis 113: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Agitation, Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0036, MMRM; LS Mean Difference = -0.38, 95% CI 2-sided [-0.63 to -0.13], Standard Error of Mean 0.126
Statistical Analysis 114: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Agitation, Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0498, MMRM; LS Mean Difference = -0.26, 95% CI 2-sided [-0.52 to 0.00], Standard Error of Mean 0.131
Statistical Analysis 115: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Agitation, Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5111, MMRM; LS Mean Difference = -0.10, 95% CI 2-sided [-0.39 to 0.20], Standard Error of Mean 0.147
Statistical Analysis 116: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Agitation, Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5839, MMRM; LS Mean Difference = -0.09, 95% CI 2-sided [-0.39 to 0.22], Standard Error of Mean 0.155
Statistical Analysis 117: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Agitation, Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1905, MMRM; LS Mean Difference = -0.13, 95% CI 2-sided [-0.33 to 0.07], Standard Error of Mean 0.100
Statistical Analysis 118: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Psychic, Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1767, MMRM; LS Mean Difference = -0.22, 95% CI 2-sided [-0.54 to 0.10], Standard Error of Mean 0.162
Statistical Analysis 119: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Psychic, Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5182, MMRM; LS Mean Difference = -0.12, 95% CI 2-sided [-0.47 to 0.24], Standard Error of Mean 0.180
Statistical Analysis 120: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Psychic, Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3930, MMRM; LS Mean Difference = -0.16, 95% CI 2-sided [-0.53 to 0.21], Standard Error of Mean 0.185
Statistical Analysis 121: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Psychic, Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5212, MMRM; LS Mean Difference = -0.12, 95% CI 2-sided [-0.50 to 0.25], Standard Error of Mean 0.189
Statistical Analysis 122: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Psychic, Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4741, MMRM; LS Mean Difference = -0.13, 95% CI 2-sided [-0.50 to 0.23], Standard Error of Mean 0.184
Statistical Analysis 123: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Psychic, Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4482, MMRM; LS Mean Difference = -0.14, 95% CI 2-sided [-0.51 to 0.23], Standard Error of Mean 0.186
Statistical Analysis 124: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Psychic, Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0963, MMRM; LS Mean Difference = -0.31, 95% CI 2-sided [-0.69 to 0.06], Standard Error of Mean 0.187
Statistical Analysis 125: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Psychic, Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0030, MMRM; LS Mean Difference = -0.52, 95% CI 2-sided [-0.86 to -0.18], Standard Error of Mean 0.171
Statistical Analysis 126: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Psychic, Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1116, MMRM; LS Mean Difference = -0.28, 95% CI 2-sided [-0.63 to 0.07], Standard Error of Mean 0.177
Statistical Analysis 127: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Psychic, Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0040, MMRM; LS Mean Difference = -0.51, 95% CI 2-sided [-0.86 to -0.17], Standard Error of Mean 0.173
Statistical Analysis 128: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Psychic, Day 14 : MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.8253, MMRM; LS Mean Difference = -0.05, 95% CI 2-sided [-0.54 to 0.43], Standard Error of Mean 0.244
Statistical Analysis 129: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Psychic, Day 21 : MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5795, MMRM; LS Mean Difference = 0.12, 95% CI 2-sided [-0.30 to 0.53], Standard Error of Mean 0.209
Statistical Analysis 130: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Psychic, Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4032, MMRM; LS Mean Difference = 0.15, 95% CI 2-sided [-0.21 to 0.51], Standard Error of Mean 0.182
Statistical Analysis 131: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Somatic, Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6117, MMRM; LS Mean Difference = -0.07, 95% CI 2-sided [-0.33 to 0.20], Standard Error of Mean 0.133
Statistical Analysis 132: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Somatic, Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4716, MMRM; LS Mean Difference = -0.09, 95% CI 2-sided [-0.35 to 0.16], Standard Error of Mean 0.130
Statistical Analysis 133: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Somatic, Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6041, MMRM; LS Mean Difference = -0.07, 95% CI 2-sided [-0.34 to 0.20], Standard Error of Mean 0.136
Statistical Analysis 134: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Somatic, Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0424, MMRM; LS Mean Difference = -0.27, 95% CI 2-sided [-0.53 to -0.01], Standard Error of Mean 0.132
Statistical Analysis 135: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Somatic, Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7622, MMRM; LS Mean Difference = -0.04, 95% CI 2-sided [-0.32 to 0.23], Standard Error of Mean 0.138
Statistical Analysis 136: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Somatic, Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2689, MMRM; LS Mean Difference = -0.14, 95% CI 2-sided [-0.40 to 0.11], Standard Error of Mean 0.130
Statistical Analysis 137: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Somatic, Hour 48 : MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2110, MMRM; LS Mean Difference = -0.17, 95% CI 2-sided [-0.44 to 0.10], Standard Error of Mean 0.134
Statistical Analysis 138: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Somatic, Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5873, MMRM; LS Mean Difference = -0.07, 95% CI 2-sided [-0.34 to 0.20], Standard Error of Mean 0.135
Statistical Analysis 139: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Somatic, Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0450, MMRM; LS Mean Difference = -0.23, 95% CI 2-sided [-0.46 to -0.01], Standard Error of Mean 0.114
Statistical Analysis 140: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Somatic, Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0847, MMRM; LS Mean Difference = -0.26, 95% CI 2-sided [-0.57 to 0.04], Standard Error of Mean 0.152
Statistical Analysis 141: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Somatic, Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2522, MMRM; LS Mean Difference = 0.22, 95% CI 2-sided [-0.16 to 0.60], Standard Error of Mean 0.189
Statistical Analysis 142: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Somatic, day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5026, MMRM; LS Mean Difference = -0.11, 95% CI 2-sided [-0.43 to 0.21], Standard Error of Mean 0.160
Statistical Analysis 143: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Anxiety Somatic, Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5911, MMRM; LS Mean Difference = -0.08, 95% CI 2-sided [-0.38 to 0.22], Standard Error of Mean 0.149
Statistical Analysis 144: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms Gastrointestinal, Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5800, MMRM; LS Mean Difference = 0.07, 95% CI 2-sided [-0.18 to 0.31], Standard Error of Mean 0.122
Statistical Analysis 145: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms Gastrointestinal, Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6754, MMRM; LS Mean Difference = -0.05, 95% CI 2-sided [-0.31 to 0.20], Standard Error of Mean 0.129
Statistical Analysis 146: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms Gastrointestinal, Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1006, MMRM; LS Mean Difference = 0.19, 95% CI 2-sided [-0.04 to 0.42], Standard Error of Mean 0.116
Statistical Analysis 147: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms Gastrointestinal, Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3588, MMRM; LS Mean Difference = 0.11, 95% CI 2-sided [-0.13 to 0.35], Standard Error of Mean 0.120
Statistical Analysis 148: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms Gastrointestinal, Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5807, MMRM; LS Mean Difference = -0.06, 95% CI 2-sided [-0.28 to 0.16], Standard Error of Mean 0.109
Statistical Analysis 149: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms Gastrointestinal, Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4241, MMRM; LS Mean Difference = 0.09, 95% CI 2-sided [-0.13 to 0.31], Standard Error of Mean 0.112
Statistical Analysis 150: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms Gastrointestinal, Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7984, MMRM; LS Mean Difference = -0.03, 95% CI 2-sided [-0.26 to 0.20], Standard Error of Mean 0.115
Statistical Analysis 151: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms Gastrointestinal, Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.8732, MMRM; LS Mean Difference = 0.02, 95% CI 2-sided [-0.22 to 0.26], Standard Error of Mean 0.122
Statistical Analysis 152: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms Gastrointestinal, Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.8621, MMRM; LS Mean Difference = 0.02, 95% CI 2-sided [-0.19 to 0.23], Standard Error of Mean 0.107
Statistical Analysis 153: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms Gastrointestinal, Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1087, MMRM; LS Mean Difference = -0.20, 95% CI 2-sided [-0.45 to 0.05], Standard Error of Mean 0.126
Statistical Analysis 154: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms Gastrointestinal, Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2153, MMRM; LS Mean Difference = -0.16, 95% CI 2-sided [-0.41 to 0.09], Standard Error of Mean 0.125
Statistical Analysis 155: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms Gastrointestinal, Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1422, MMRM; LS Mean Difference = -0.22, 95% CI 2-sided [-0.51 to 0.07], Standard Error of Mean 0.145
Statistical Analysis 156: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms Gastrointestinal, Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7211, MMRM; LS Mean Difference = 0.04, 95% CI 2-sided [-0.19 to 0.27], Standard Error of Mean 0.114
Statistical Analysis 157: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms General, Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.8224, MMRM; LS Mean Difference = 0.02, 95% CI 2-sided [-0.18 to 0.23], Standard Error of Mean 0.103
Statistical Analysis 158: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms General, Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6362, MMRM; LS Mean Difference = -0.06, 95% CI 2-sided [-0.31 to 0.19], Standard Error of Mean 0.126
Statistical Analysis 159: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms General, Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6094, MMRM; LS Mean Difference = -0.06, 95% CI 2-sided [-0.31 to 0.18], Standard Error of Mean 0.123
Statistical Analysis 160: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms General, Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0457, MMRM; LS Mean Difference = -0.25, 95% CI 2-sided [-0.49 to 0.00], Standard Error of Mean 0.123
Statistical Analysis 161: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms General, Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5691, MMRM; LS Mean Difference = -0.08, 95% CI 2-sided [-0.36 to 0.20], Standard Error of Mean 0.140
Statistical Analysis 162: Comparison: Placebo; Somatic Symptoms General, Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2942, MMRM; LS Mean Difference = -0.14, 95% CI 2-sided [-0.40 to 0.12], Standard Error of Mean 0.130
Statistical Analysis 163: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms General, Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5389, MMRM; LS Mean Difference = -0.08, 95% CI 2-sided [-0.35 to 0.19], Standard Error of Mean 0.136
Statistical Analysis 164: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms General, Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4061, MMRM; LS Mean Difference = -0.12, 95% CI 2-sided [-0.40 to 0.16], Standard Error of Mean 0.141
Statistical Analysis 165: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms General, Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0990, MMRM; LS Mean Difference = -0.25, 95% CI 2-sided [-0.56 to 0.05], Standard Error of Mean 0.153
Statistical Analysis 166: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms General, Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0108, MMRM; LS Mean Difference = -0.36, 95% CI 2-sided [-0.63 to -0.08], Standard Error of Mean 0.138
Statistical Analysis 167: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms General, Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0889, MMRM; LS Mean Difference = -0.28, 95% CI 2-sided [-0.59 to 0.04], Standard Error of Mean 0.160
Statistical Analysis 168: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms General, Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3721, MMRM; LS Mean Difference = 0.15, 95% CI 2-sided [-0.18 to 0.49], Standard Error of Mean 0.169
Statistical Analysis 169: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Somatic Symptoms General, Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5513, MMRM; LS Mean Difference = -0.08, 95% CI 2-sided [-0.36 to 0.20], Standard Error of Mean 0.141
Statistical Analysis 170: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Genital Symptoms, Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0748, MMRM; LS Mean Difference = 0.12, 95% CI 2-sided [-0.01 to 0.26], Standard Error of Mean 0.067
Statistical Analysis 171: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Genital Symptoms, Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3545, MMRM; LS Mean Difference = 0.08, 95% CI 2-sided [-0.09 to 0.25], Standard Error of Mean 0.087
Statistical Analysis 172: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Genital Symptoms, Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6531, MMRM; LS Mean Difference = 0.04, 95% CI 2-sided [-0.14 to 0.23], Standard Error of Mean 0.094
Statistical Analysis 173: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Genital Symptoms, Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7520, MMRM; LS Mean Difference = -0.04, 95% CI 2-sided [-0.26 to 0.19], Standard Error of Mean 0.115
Statistical Analysis 174: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Genital Symptoms, Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.8861, MMRM; LS Mean Difference = -0.02, 95% CI 2-sided [-0.26 to 0.23], Standard Error of Mean 0.123
Statistical Analysis 175: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Genital Symptoms, Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3280, MMRM; LS Mean Difference = -0.12, 95% CI 2-sided [-0.38 to 0.13], Standard Error of Mean 0.127
Statistical Analysis 176: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Genital Symptoms, Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1123, MMRM; LS Mean Difference = -0.21, 95% CI 2-sided [-0.46 to 0.05], Standard Error of Mean 0.128
Statistical Analysis 177: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Genital Symptoms, Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2541, MMRM; LS Mean Difference = -0.13, 95% CI 2-sided [-0.36 to 0.10], Standard Error of Mean 0.116
Statistical Analysis 178: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Genital Symptoms, Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0110, MMRM; LS Mean Difference = -0.37, 95% CI 2-sided [-0.66 to -0.09], Standard Error of Mean 0.143
Statistical Analysis 179: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Genital Symptoms, Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7720, MMRM; LS Mean Difference = -0.05, 95% CI 2-sided [-0.36 to 0.27], Standard Error of Mean 0.158
Statistical Analysis 180: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Genital Symptoms, Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6311, MMRM; LS Mean Difference = -0.10, 95% CI 2-sided [-0.52 to 0.32], Standard Error of Mean 0.210
Statistical Analysis 181: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Genital Symptoms, Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6877, MMRM; LS Mean Difference = -0.08, 95% CI 2-sided [-0.50 to 0.33], Standard Error of Mean 0.207
Statistical Analysis 182: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Genital Symptoms, Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2465, MMRM; LS Mean Difference = 0.22, 95% CI 2-sided [-0.15 to 0.58], Standard Error of Mean 0.186
Statistical Analysis 183: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Hypochondriasis, Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1279, MMRM; LS Mean Difference = -0.16, 95% CI 2-sided [-0.36 to 0.05], Standard Error of Mean 0.101
Statistical Analysis 184: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Hypochondriasis, Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3946, MMRM; LS Mean Difference = -0.08, 95% CI 2-sided [-0.26 to 0.10], Standard Error of Mean 0.093
Statistical Analysis 185: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Hypochondriasis, Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6694, MMRM; LS Mean Difference = -0.04, 95% CI 2-sided [-0.23 to 0.15], Standard Error of Mean 0.095
Statistical Analysis 186: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Hypochondriasis, Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1113, MMRM; LS Mean Difference = -0.16, 95% CI 2-sided [-0.36 to 0.04], Standard Error of Mean 0.100
Statistical Analysis 187: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Hypochondriasis, Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5811, MMRM; LS Mean Difference = 0.05, 95% CI 2-sided [-0.13 to 0.23], Standard Error of Mean 0.089
Statistical Analysis 188: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Hypochondriasis, Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6794, MMRM; LS Mean Difference = -0.04, 95% CI 2-sided [-0.25 to 0.17], Standard Error of Mean 0.106
Statistical Analysis 189: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Hypochondriasis, Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6031, MMRM; LS Mean Difference = 0.05, 95% CI 2-sided [-0.14 to 0.25], Standard Error of Mean 0.099
Statistical Analysis 190: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Hypochondriasis, Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6673, MMRM; LS Mean Difference = -0.04, 95% CI 2-sided [-0.24 to 0.15], Standard Error of Mean 0.099
Statistical Analysis 191: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Hypochondriasis, Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6472, MMRM; LS Mean Difference = -0.05, 95% CI 2-sided [-0.25 to 0.16], Standard Error of Mean 0.102
Statistical Analysis 192: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Hypochondriasis, Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.8654, MMRM; LS Mean Difference = -0.02, 95% CI 2-sided [-0.26 to 0.22], Standard Error of Mean 0.119
Statistical Analysis 193: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Hypochondriasis, Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2101, MMRM; LS Mean Difference = -0.18, 95% CI 2-sided [-0.48 to 0.11], Standard Error of Mean 0.140
Statistical Analysis 194: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Hypochondriasis, Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7128, MMRM; LS Mean Difference = -0.05, 95% CI 2-sided [-0.30 to 0.21], Standard Error of Mean 0.126
Statistical Analysis 195: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Hypochondriasis, Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3297, MMRM; LS Mean Difference = -0.09, 95% CI 2-sided [-0.27 to 0.09], Standard Error of Mean 0.090
Statistical Analysis 196: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Loss of weight, Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4493, MMRM; LS Mean Difference = 0.05, 95% CI 2-sided [-0.08 to 0.19], Standard Error of Mean 0.069
Statistical Analysis 197: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Loss of weight, Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0717, MMRM; LS Mean Difference = 0.15, 95% CI 2-sided [-0.01 to 0.31], Standard Error of Mean 0.081
Statistical Analysis 198: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Loss of Weight, Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1054, MMRM; LS Mean Difference = 0.11, 95% CI 2-sided [-0.02 to 0.24], Standard Error of Mean 0.066
Statistical Analysis 199: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Loss of Weight, Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0408, MMRM; LS Mean Difference = 0.18, 95% CI 2-sided [0.01 to 0.36], Standard Error of Mean 0.088
Statistical Analysis 200: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Loss of Weight, Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0233, MMRM; LS Mean Difference = 0.20, 95% CI 2-sided [0.03 to 0.38], Standard Error of Mean 0.088
Statistical Analysis 201: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Loss of Weight, Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3610, MMRM; LS Mean Difference = 0.08, 95% CI 2-sided [-0.09 to 0.26], Standard Error of Mean 0.088
Statistical Analysis 202: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Loss of Weight, Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2358, MMRM; LS Mean Difference = 0.12, 95% CI 2-sided [-0.08 to 0.32], Standard Error of Mean 0.100
Statistical Analysis 203: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Loss of Weight, Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9492, MMRM; LS Mean Difference = 0.01, 95% CI 2-sided [-0.16 to 0.17], Standard Error of Mean 0.085
Statistical Analysis 204: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Loss of Weight, Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4352, MMRM; LS Mean Difference = -0.08, 95% CI 2-sided [-0.28 to 0.12], Standard Error of Mean 0.102
Statistical Analysis 205: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Loss of Weight, Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1176, MMRM; LS Mean Difference = 0.20, 95% CI 2-sided [-0.05 to 0.44], Standard Error of Mean 0.125
Statistical Analysis 206: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Loss of Weight, Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7812, MMRM; LS Mean Difference = 0.05, 95% CI 2-sided [-0.30 to 0.40], Standard Error of Mean 0.174
Statistical Analysis 207: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Loss of Weight, Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.5085, MMRM; LS Mean Difference = -0.12, 95% CI 2-sided [-0.48 to 0.24], Standard Error of Mean 0.182
Statistical Analysis 208: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Loss of Weight, Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.8274, MMRM; LS Mean Difference = 0.03, 95% CI 2-sided [-0.28 to 0.34], Standard Error of Mean 0.156
Statistical Analysis 209: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insight, Hour 2: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3675, MMRM; LS Mean Difference = -0.04, 95% CI 2-sided [-0.13 to 0.05], Standard Error of Mean 0.045
Statistical Analysis 210: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insight, Hour 4: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1818, MMRM; LS Mean Difference = -0.06, 95% CI 2-sided [-0.15 to 0.03], Standard Error of Mean 0.045
Statistical Analysis 211: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insight, Hour 8: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0826, MMRM; LS Mean Difference = -0.08, 95% CI 2-sided [-0.17 to 0.01], Standard Error of Mean 0.045
Statistical Analysis 212: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insight, Hour 12: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6436, MMRM; LS Mean Difference = -0.02, 95% CI 2-sided [-0.11 to 0.07], Standard Error of Mean 0.045
Statistical Analysis 213: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insight, Hour 24: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1827, MMRM; LS Mean Difference = -0.06, 95% CI 2-sided [-0.15 to 0.03], Standard Error of Mean 0.045
Statistical Analysis 214: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insight, Hour 36: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9859, MMRM; LS Mean Difference = 0.00, 95% CI 2-sided [-0.09 to 0.09], Standard Error of Mean 0.045
Statistical Analysis 215: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insight, Hour 48: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6672, MMRM; LS Mean Difference = 0.02, 95% CI 2-sided [-0.07 to 0.11], Standard Error of Mean 0.045
Statistical Analysis 216: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insight, Hour 60: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2031, MMRM; LS Mean Difference = 0.06, 95% CI 2-sided [-0.03 to 0.15], Standard Error of Mean 0.046
Statistical Analysis 217: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insight, Hour 72: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6664, MMRM; LS Mean Difference = 0.02, 95% CI 2-sided [-0.07 to 0.11], Standard Error of Mean 0.045
Statistical Analysis 218: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insight, Day 7: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.3417, MMRM; LS Mean Difference = -0.04, 95% CI 2-sided [-0.13 to 0.05], Standard Error of Mean 0.045
Statistical Analysis 219: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insight, Day 14: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.6622, MMRM; LS Mean Difference = -0.02, 95% CI 2-sided [-0.12 to 0.08], Standard Error of Mean 0.051
Statistical Analysis 220: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insight, Day 21: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9087, MMRM; LS Mean Difference = -0.01, 95% CI 2-sided [-0.11 to 0.09], Standard Error of Mean 0.051
Statistical Analysis 221: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Insight, Day 30: MMRM was used for analysis. The change from baseline in HAM-D individual item score at each visit was the dependent variable. Treatment, baseline HAM-D individual item score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms were explanatory variables included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.8263, MMRM; LS Mean Difference = 0.01, 95% CI 2-sided [-0.08 to 0.10], Standard Error of Mean 0.046

8. Secondary Outcome: Change From Baseline at Key Time Points in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in participants with mood disorders. It was designed as an adjunct to the HAM-D, to be more sensitive than the Hamilton Scale to the changes brought on by antidepressants and other forms of treatment. Each item yielded a score of 0 to 6. The MADRS total score was calculated as the sum of the 10 individual item scores, which ranged from 0 to 60. Higher MADRS scores indicates more severe depression. A negative change from baseline indicates less severe depression. A positive change from baseline indicates more severe depression.
Time Frame: Baseline, Hour 60, Days 7 and 30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 53 | 51
score on a scale
  Hour 60: number analyzed (Participants) | 52 | 49
  Hour 60 | -15.66 (1.329) | -20.52 (1.333)
  Day 7: number analyzed (Participants) | 53 | 49
  Day 7 | -15.35 (1.658) | -18.91 (1.676)
  Day 30: number analyzed (Participants) | 52 | 48
  Day 30 | -20.52 (1.489) | -20.48 (1.504)
Statistical Analysis 1: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Hour 60: MMRM was used for analysis. The change from baseline in MADRS total score at each visit was the dependent variable. Treatment, baseline MADRS total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.0033, MMRM; LS mean difference = -4.86, 95% CI 2-sided [-8.06 to -1.66], Standard Error of Mean 1.612
Statistical Analysis 2: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Day 7: MMRM was used for analysis. The change from baseline in MADRS total score at each visit was the dependent variable. Treatment, baseline MADRS total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1017, MMRM; LS mean difference = -3.56, 95% CI 2-sided [-7.84 to 0.72], Standard Error of Mean 2.154
Statistical Analysis 3: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Day 30: MMRM was used for analysis. The change from baseline in MADRS total score at each visit was the dependent variable. Treatment, baseline MADRS total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.9845, MMRM; LS mean difference = 0.04, 95% CI 2-sided [-3.72 to 3.79], Standard Error of Mean 1.884

9. Secondary Outcome: Percentage of Participants With Clinical Global Impression - Improvement (CGI-I) Response
Description: The CGI-I response was defined as having a score of 1 (very much improved) or 2 (much improved). CGI-I item employs a 7-point Likert scale to measure the overall improvement in the participant's condition post-treatment. The investigator rated the participant's total improvement whether or not it was due entirely to drug treatment. Response choices include: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. The CGI-I was only rated at post-treatment assessments. By definition, all CGI-I assessments were evaluated against baseline conditions.
Time Frame: Hour 60, Days 7 and 30
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 53 | 51
percentage of participants
  Hour 60: number analyzed (Participants) | 52 | 49
  Hour 60 | 55.8 | 79.6
  Day 7: number analyzed (Participants) | 53 | 50
  Day 7 | 54.7 | 70.0
  Day 30: number analyzed (Participants) | 52 | 48
  Day 30 | 78.8 | 81.3
Statistical Analysis 1: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Hour 60: GEE method was used for analysis. CGI-I response at each visit was the dependent variable. Treatment, baseline CGI-S score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model; Test type: Superiority; p = 0.0005, GEE method; Odds Ratio (OR) = 5.0, 95% CI 2-sided [2.0 to 12.5]
Statistical Analysis 2: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Day 7: GEE method was used for analysis. CGI-I response at each visit was the dependent variable. Treatment, baseline CGI-S score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model; Test type: Superiority; p = 0.0478, GEE method; Odds Ratio (OR) = 2.9, 95% CI 2-sided [1.0 to 8.4]
Statistical Analysis 3: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Day 30: GEE method was used for analysis. CGI-I response at each visit was the dependent variable. Treatment, baseline CGI-S score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model; Test type: Superiority; p = 0.4399, GEE method; Odds Ratio (OR) = 1.5, 95% CI 2-sided [0.5 to 4.6]

10. Secondary Outcome: Change From Baseline in the Generalized Anxiety Disorder 7-Item Scale (GAD-7) Total Score
Description: The GAD-7 is a participant-rated, generalized anxiety symptom severity scale. Scoring for GAD-7 generalized anxiety is calculated by assigning scores of 0 = "not at all sure," 1 = "several days," 2 = "over half the days," and 3 = "nearly every day" to the response categories. The GAD-7 total score for the seven items ranges from 0 to 21, where a score of 0 to 4 = minimal anxiety, 5 to 9 = mild anxiety, 10 to 14 = moderate anxiety, and 15 to 21 = severe anxiety. The GAD-7 total score was calculated as the sum of the seven individual item scores. A negative change from baseline indicates less anxiety. A positive change from baseline indicates more anxiety.
Time Frame: Baseline, Hour 60, Days 7, 14, 21 and 30
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 53 | 51
score on a scale
  Hour 60: number analyzed (Participants) | 51 | 46
  Hour 60 | -6.41 (0.814) | -7.58 (0.850)
  Day 7: number analyzed (Participants) | 51 | 48
  Day 7 | -7.67 (0.858) | -8.43 (0.879)
  Day 14: number analyzed (Participants) | 31 | 29
  Day 14 | -7.90 (0.937) | -9.76 (0.961)
  Day 21: number analyzed (Participants) | 31 | 30
  Day 21 | -8.92 (1.053) | -10.88 (1.081)
  Day 30: number analyzed (Participants) | 50 | 46
  Day 30 | -9.89 (0.884) | -10.20 (0.913)
Statistical Analysis 1: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Hour 60: MMRM was used for the analysis. The change from baseline in GAD-7 total score at each visit was the dependent variable. Treatment, baseline GAD-7 total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.2636, MMRM; LS Mean Difference = -1.17, 95% CI 2-sided [-3.24 to 0.90], Standard Error of Mean 1.041
Statistical Analysis 2: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Day 7: MMRM was used for the analysis. The change from baseline in GAD-7 total score at each visit was the dependent variable. Treatment, baseline GAD-7 total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.4897, MMRM; LS Mean Difference = -0.76, 95% CI 2-sided [-2.96 to 1.43], Standard Error of Mean 1.103
Statistical Analysis 3: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Day 14: MMRM was used for the analysis. The change from baseline in GAD-7 total score at each visit was the dependent variable. Treatment, baseline GAD-7 total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1341, MMRM; LS Mean Difference = -1.86, 95% CI 2-sided [-4.30 to 0.59], Standard Error of Mean 1.227
Statistical Analysis 4: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Day 21: MMRM was used for the analysis. The change from baseline in GAD-7 total score at each visit was the dependent variable. Treatment, baseline GAD-7 total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.1691, MMRM; LS Mean Difference = -1.95, 95% CI 2-sided [-4.76 to 0.85], Standard Error of Mean 1.408
Statistical Analysis 5: Comparison: Placebo vs SAGE-547 90 μg/kg/h; Change at Day 30: MMRM was used for the analysis. The change from baseline in GAD-7 total score at each visit was the dependent variable. Treatment, baseline GAD-7 total score, pooled center, baseline antidepressant use, visit time point, and visit time point-by-treatment interaction terms as explanatory variables were included in the model. All explanatory variables including pooled center were treated as fixed effects; Test type: Superiority; p = 0.7852, MMRM; LS Mean Difference = -0.31, 95% CI 2-sided [-2.60 to 1.97], Standard Error of Mean 1.149

11. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Event (TEAE)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an AE with onset on or after the start of study drug infusion, or any worsening of a pre-existing medical condition/AE with onset on or after the start of study drug infusion.
Time Frame: Up to approximately 37 days
Population: The safety set included all randomized participants who started the study drug infusion.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 53 | 51
percentage of participants | 45.3 | 49.0

12. Secondary Outcome: Time to Change in Antidepressant Medication
Description: The time to first start or increase in the dose and time to first stop or decrease in the dose of any antidepressant medication.
Time Frame: Up to approximately 37 days
Population: as for outcome 3
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | SAGE-547 90 μg/kg/h
Number analyzed (Participants) | 53 | 51
days
  Time to first start/increase in dose: number analyzed (Participants) | 7 | 5
  Time to first start/increase in dose | 8 [4 to 13] | 10 [7 to 17]
  Time to first stop/decrease in dose: number analyzed (Participants) | 0 | 1
  Time to first stop/decrease in dose |  | 18 [18 to 18]

ADVERSE EVENTS:
Time Frame: Up to approximately 37 days
Description: The Safety Set included all randomized participants who started the study drug infusion.
Arm/Group | Placebo | SAGE-547 90 μg/kg/h
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/53 | 1/51
Other Adverse Events (participants affected / at risk) | 13/53 | 21/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=53) | SAGE-547 90 μg/kg/h (N=51)
Altered state of consciousness (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=53) | SAGE-547 90 μg/kg/h (N=51)
Nausea (Gastrointestinal disorders) | 2 | 5
Fatigue (General disorders) | 2 | 3
Infusion site pain (General disorders) | 2 | 5
Dizziness (Nervous system disorders) | 4 | 5
Headache (Nervous system disorders) | 6 | 9
Somnolence (Nervous system disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).

DOCUMENTS (2):
  • Study Protocol (2017-03-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT02942017/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/17/NCT02942017/SAP_001.pdf